# Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest – A Randomized, Double-Blind, Placebo-Controlled Trial

Acronym: VAM-IHCA

# TRIAL PROTOCOL

Version 1.8 Oct 30, 2020

EudraCT number: 2017-004773-13

ClinicalTrials.gov number: NCT03640949

Principal investigator and sponsor:

Lars W. Andersen, M.D., M.P.H., Ph.D., D.M.Sc.

**Associate Professor** 

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Palle Juul Jensens Boulevard 99, Bygning J, Plan 1

8200 Aarhus N, Denmark

Phone: +4551781511

Email: lwandersen@clin.au.dk

VAM-IHCA Protocol – version 1.8 Page **1** of **80** 

# Content

| Preface | 6 |
|-------------------------------------------------------------|----|
| List of abbreviations | 7 |
| Overview | 8 |
| Trial flow chart | 9 |
| Steering committee | 10 |
| Trial sites | 12 |
| Pharmacy | 14 |
| Amendments | 15 |
| 1. BACKGROUND | 19 |
| 1.1 In-hospital cardiac arrest | 19 |
| 1.1.1 Incidence and mortality | 19 |
| 1.1.2 An understudied entity | 19 |
| 1.1.3 Pathophysiology | 19 |
| 1.2 Vasopressin | 20 |
| 1.2.1 Pharmacology | 20 |
| 1.2.2 Use outside cardiac arrest | 20 |
| 1.2.3 Use in cardiac arrest | 20 |
| 1.3 Methylprednisolone | 21 |
| 1.3.1 Pharmacology | 21 |
| 1.3.2 Use outside cardiac arrest | 21 |
| 1.3.3 Use in cardiac arrest | 21 |
| 1.4 The vasopressin, steroids, and epinephrine (VSE) trials | 22 |
| 1.5 Guidelines regarding vasopressin and glucocorticoids | 22 |
| 1.6 Standard of care | 23 |
| 1.7 Post-cardiac arrest glucocorticoids | 23 |
| 2. TRIAL OBJECTIVES AND HYPOTHESES | 24 |
| 3. TRIAL DESIGN | 25 |
| 3.1 Overview | 25 |
| 3.2 Allocation | 25 |
| 3.3 Interventions | 25 |
| 3.3.1 Methylprednisolone and vasopressin | 25 |
| 3.3.2 Placebo | 25 |

| 3.3.3 Procedures | 26 |
|-------------------------------------------------------------|----|
| 3.3.4 Overview of study medication | 26 |
| 3.4 Blinding | 27 |
| 3.5 Trial procedures | 27 |
| 3.5.1 Patients | 27 |
| 3.5.2 Clinical personnel | 28 |
| 4. SETTING AND PATIENT POPULATION | 28 |
| 4.1 Setting | 28 |
| 4.2 Inclusion criteria | 28 |
| 4.3 Exclusion criteria | 28 |
| 4.4 Co-enrollment | 29 |
| 5. OUTCOMES | 29 |
| 5.1 Primary outcome | 29 |
| 5.1.1 Definition | 29 |
| 5.1.2 Rationale | 30 |
| 5.2 Secondary outcomes | 30 |
| 5.2.1 Definitions | 30 |
| 5.2.2 Rationale | 31 |
| 5.3 Tertiary outcomes | 31 |
| 5.4 Harm | 33 |
| 5.4.1 General consideration | 33 |
| 5.4.2 Definitions | 33 |
| 5.4.3 Specific adverse events | 34 |
| 5.4.4 Timeline | 35 |
| 5.4.5 Suspected Unexpected Serious Adverse Reaction (SUSAR) | 35 |
| 5.5 Additional follow-up | 35 |
| 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN | 36 |
| 6.1 Sample size calculation | 36 |
| 6.2 Statistical analysis plan | 37 |
| 6.2.1 General considerations | 37 |
| 6.2.2 Primary and secondary outcomes | 37 |
| 6.2.3 Subgroup analyses | 37 |
| 6.2.4 Addition analyses and outcomes | 38 |
| 6.2.5 Missing data | 38 |

| 6.2.6 Multiple comparisons | 38 |
|----------------------------------------------------|----|
| 6.2.7 Statistical stopping criteria | 39 |
| 7. DATA COLLECTION AND MANAGEMENT | 39 |
| 7.1 Data collection process | 39 |
| 7.2 Variables | 39 |
| 7.2.1 Overview | 39 |
| 7.2.2 Pre-cardiac arrest characteristics | 40 |
| 7.2.3 Cardiac arrest characteristics | 41 |
| 7.2.3 Post-cardiac arrest characteristics | 41 |
| 7.2.4 Outcomes | 42 |
| 7.3 Data quality and validity | 42 |
| 7.4 Data storage and security | 42 |
| 7.5 Data access | 43 |
| 7.6 DANARREST | 43 |
| 8. CLINICAL TREATMENT | 43 |
| 9. ETHICAL CONSIDERATIONS | 43 |
| 9.1 Clinical equipoise | 43 |
| 9.1.1 Potential benefits | 43 |
| 9.1.2 Potential harms | 44 |
| 9.1.3 Risk/benefit ratio | 44 |
| 9.2 Research in cardiac arrest | 44 |
| 9.2.1 General considerations | 44 |
| 9.2.2 Danish regulations | 45 |
| 9.2.3 Regulations in relation to the current trial | 46 |
| 9.3 Procedures | 46 |
| 9.3.1 Ethical review committee | 46 |
| 9.3.2 Trial-specific procedures | 47 |
| 9.3.3 Insurance | 47 |
| 10. MONITORING | 47 |
| 10.1 Good Clinical Practice monitoring | 47 |
| 10.2 Independent data-monitoring committee (IDMC) | 48 |
| 11. TIMELINE AND ENROLLMENT | 49 |
| 11.1 Timeline | 49 |
| 11.2 Feasibility | 50 |

| | 11.3 Enrollment | 50 |
|---|---|---|
| | 11.4 Additional sites | 51 |
| 12 | PUBLICATION PLAN | 51 |
| 13 | 3. DATA SHARING | 51 |
| 14 | I. FUNDING | 52 |
| 15 | i. TASKS AND RESPONSIBILITIES | 52 |
| Re | eferences | 53 |
| Αį | ppendices | 64 |
| | Appendix 1: Conflict of interest disclosures for the steering committee members | 64 |
| | Appendix 2: Study kit and drug labeling (Danish) | 70 |
| | Appendix 3: Draft of CONSORT flow diagram | 71 |
| | Appendix 4: Case report form (Danish) | 72 |
| | Appendix 5: DANARREST case report form (Danish) | . 73 |
| | Appendix 6: Charter for the independent data-monitoring committee (IDMC) | . 75 |

#### **Preface**

The "Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest – A Randomized, Double-Blind, Placebo-Controlled Trial" (VAM-IHCA) will be conducted according to this protocol. The trial will be conducted in accordance with all applicable national and international laws, regulations, and guidelines including the revised version of the Declaration of Helsinki¹, European regulations², and the international Good Clinical Practice guidelines³. The trial and this protocol is developed in accordance with the International Conference on Harmonization (ICH) guidelines³-5 and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) statement<sup>6,7</sup>. The principal investigator wrote the protocol with input from the steering committee. Any substantial changes or amendments to the protocol will be clearly documented and communicated to all relevant parties.

30/10 - 2020

Date

Lars W. Andersen, M.D., M.P.H., Ph.D., D.M.Sc.

as W. Ander

# **List of abbreviations**

CPC: Cerebral performance category

CPR: Cardiopulmonary resuscitation

ICH: International Conference on Harmonization

IDMC: Independent data-monitoring committee

IHCA: In-hospital cardiac arrest

ILCOR: International Liaison Committee on Resuscitation

mRS: Modified Rankin scale

OHCA: Out-of-hospital cardiac arrest

ROSC: Return of spontaneous circulation

SOFA: Sequential organ failure assessment

SPIRIT: Standard Protocol Items: Recommendations for Interventional Trials

VSE: Vasopressin, steroids, and epinephrine

# Overview

| Registry and trial number | EudraCT number: 2017-004773-13, ClinicalTrials.gov number: NCT03640949 | |
|---|---|---|
| Date of registration | EudraCT: 25/1-2018, ClinicalTrials.gov: 21/8-2018 | |
| Sources of monetary or | Aarhus University Research Foundation | |
| material support | Department of Clinical Medicine, Aarhus University | |
| | Independent Research Fund Denmark | |
| | Amomed Pharma GmbH (only vasopressin) | |
| Primary sponsor | Lars W. Andersen, Aarhus University | |
| Contact | Lars W. Andersen, lwandersen@clin.au.dk | |
| Title | Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest – A<br>Randomized, Double-Blind, Placebo-Controlled Trial | |
| Country of recruitment | Denmark | |
| Condition studied | In-hospital cardiac arrest | |
| Interventions | Methylprednisolone (40 mg) combined with | |
| | Vasopressin (20 IU per adrenaline dose, maximum 80 IU) | |
| Comparator | Placebo (for both methylprednisolone and vasopressin) | |
| Inclusion criteria | 1) In-hospital cardiac arrest | |
| | 2) Age ≥ 18 years | |
| | Received at least one dose of adrenaline during CPR | |
| Exclusion criteria | 1) Clearly documented "do-not-resuscitate" order prior to the cardiac ar | |
| | • | rior enrollment in the trial nvasive mechanical circulatory support at the time of the cardiac arrest |
| | 4) Known or suspected pregnancy at the time of the cardiac arrest | |
| Study type | Interventional | Allocation: Randomized (1:1) |
| | Intervention model: Parallel group | Masking: Double-blind |
| Date of first screening | Sept. 17, 2018 | |
| Target sample size | 492 | |
| Recruitment status | Recruiting | |
| Primary outcomes | Return of spontaneous circulation | |
| Key secondary outcomes | Survival at 30 days | |
| | Survival at 30 days with a favorable neur performance category 1 or 2) | ological outcome (cerebral |

# **Trial flow chart**



# Steering committee

Lars W. Andersen, M.D., M.P.H., Ph.D., D.M.Sc.

**Associate Professor** 

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Michael Donnino, M.D.

Director, Professor

Center for Resuscitation Science

Beth Israel Deaconess Medical Center

Harvard Medical School

Hans Kirkegaard, M.D., Ph.D., D.M.Sc.

Director, Professor

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Tobias Kurth, M.D., Sc.D.

Director, Professor

Institute of Public Health

Charité Universitätsmedizin Berlin

Bodil S. Rasmussen, M.D., Ph.D.

Professor

Department of Anesthesiology and Intensive Care

Medicine, Aalborg University Hospital

Department of Clinical Medicine, Aalborg University

Jesper Kjærgaard, M.D., Ph.D., D.M.Sc.

**Department of Cardiology** 

Rigshospitalet

Copenhagen University Hospital

Bo Løfgren, M.D., Ph.D.

Professor

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Dan Isbye, M.D., Ph.D.

Clinical Associate Professor

Department of Anesthesiology

Copenhagen University Hospital - Rigshospitalet

Jacob Moesgaard Larsen, M.D., Ph.D.

Department of Cardiology

**Aalborg University Hospital** 

Asger Granfeldt, M.D., Ph.D., D.M.Sc.

Associate Professor

Department of Anesthesiology

Aarhus University Hospital

Stine Thorhauge Zwisler, M.D., Ph.D.

Department of Anesthesiology

**Odense University Hospital** 

Søren Darling, M.D.

Department of Anesthesiology

**Odense University Hospital** 

Kasper Glerup Lauridsen, M.D.

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Kim B. Pælestik, M.D.

Department of Anesthesiology

Viborg Regional Hospital

Christoffer Sølling, M.D., Ph.D.

Department of Anesthesiology

Viborg Regional Hospital

Anders Kjærgaard, M.D., Ph.D.

Department of Anesthesiology

Horsens Regional Hospital

Dorte Due-Rasmussen, M.D.

Department of Anesthesiology

Horsens Regional Hospital

Martin Schultz, M.D., Ph.D.

Department of Internal Medicine

Copenhagen University Hospital – Herlev

Fredrik Folke, M.D., Ph.D.

Professor

Department of Cardiology

Copenhagen University Hospital – Gentofte

Kasper Iversen, M.D., D.M.Sc.

Professor

Department of Cardiology

Copenhagen University Hospital - Herlev

Mette Gitz Charlot, M.D., Ph.D.

Department of Cardiology

Copenhagen University Hospital – Gentofte

Sebastian Wiberg, M.D., Ph.D.

Department of Anesthesiology

Zealand University Hospital - Køge

Mathias Holmberg, M.D., M.P.H, Ph.D.

Research Center for Emergency Medicine

Department of Clinical Medicine

Aarhus University and Aarhus University Hospital

Rikke Malene Jepsen, M.D., Ph.D.

Department of Anesthesiology

Zealand University Hospital - Køge

#### **Conflicts of interest**

The members of the steering committee have no conflicts of interest related to the current trial. A list of all conflict of interests is provided in Appendix 1.

#### **Trial sites**

# Aarhus University Hospital - Skejby

Palle Juul-Jensens Boulevard 99

8200 Aarhus N

Denmark

Site investigator: Asger Granfeldt, granfeldt@clin.au.dk

# Aalborg University Hospital - South

Hobrovej 18 – 22

9000 Aalborg

Denmark

Site investigator: Jacob Moesgaard Larsen, jaml@rn.dk

# **Randers Regional Hospital**

Skovlyvej 15

8930 Randers NØ

Denmark

Site investigator: Kasper Glerup Lauridsen, kglerup@clin.au.dk

# Copenhagen University Hospital - Rigshospitalet

Blegdamsvej 9

2100 Copenhagen

Denmark

Site investigator: Dan Isbye, dan.lou.isbye@regionh.dk

# **Odense University Hospital**

J. B. Winsløws Vej 4

5000 Odense C

Denmark

Site investigator: Søren Darling, sorendarling@gmail.com

# **Horsens Regional Hospital**

Sundvej 30

8700 Horsens

Denmark

Site investigator: Anders Kjærgaard, andekjae@rm.dk

# **Viborg Regional Hospital**

Heibergs Alle 4

8800 Viborg

Denmark

Site investigator: Christoffer Sølling, chrsoell@rm.dk

# Copenhagen University Hospital - Gentofte

Kildegårdsvej 28

2900 Hellerup

Denmark

Site investigator: Fredrik Folke, fredrik.folke@regionh.dk

# Copenhagen University Hospital - Herlev

Herlev Ringvej 75

2730 Herlev

Denmark

Site investigator: Kasper Iversen, Kasper.Karmark.Iversen@regionh.dk

# Zealand University Hospital - Køge

Lykkebækvej 1

4600 Køge

Denmark

Site investigator: Rikke Malene Jepsen, rimj@regionsjaelland.dk

# **Pharmacy**

Skanderborg Pharmacy

Adelgade 27

8660 Skanderborg

Denmark

Contact: Heidi Svith, hei@skanderborg-apotek.dk

#### **Amendments**

#### Version 1.7 (May 14, 2020) to 1.8 (Oct. 30, 2020)

- Corrections of minor typos and grammatical issues as well as minor clarifications
- Minor change to the publication plan (section 12)
- Removal of three sites including site investigators (multiple sections)
- Multiple changes to the statistical analyses plan including (section 6):
  - Change of the primary analysis
  - Addition of a sensitivity analysis for the primary outcome
  - Subgroup analyses on both the relative and absolute scale
  - Only reporting P values for certain key outcomes
  - Removal of two subgroup analyses and addition of two
  - Analysis of survival to 90 days as a binary outcome

# Version 1.6 (Nov. 11, 2019) to 1.7 (May 14, 2020)

- Addition of four new sites (multiple sections)
- Change of site investigator in Viborg from Therese Straarup to Kim B. Pælestik (multiple sections)
- Addition of Mathias Holmberg to the steering committee (multiple sections)
- Corrections of minor typos and grammatical issues

# Version 1.5 (Apr. 4, 2019) to 1.6 (Nov. 11, 2019)

- Change of site investigator in Aalborg from Signe Juul Riddersholm to Jacob Moesgaard Larsen (multiple sections)
- Addition of a subgroup analysis based on time from adrenaline administration to first study drug and removal of the site subgroup analysis (section 6.2.3)
- Addition of funding (section 14)

# Version 1.4 (Sep. 12, 2018) to 1.5 (Apr. 4, 2019)

Addition of four sites + site investigators (multiple sections)

# Version 1.3 (Mar. 19, 2018) to 1.4 (Sep. 12, 2018)

- Corrections of minor typos and grammatical issues
- Change of address for the principal investigator (title page)

- Addition of EudraCT and ClinicalTrials.gov numbers (title page)
- Update of the overview table
- Addition of Kasper Glerup Lauridsen as a site investigator in Randers (multiple sections)
- Change of site investigator in Aalborg from Jacob Moesgaard Larsen to Signe Juul Riddersholm (multiple sections)
- Reference to Appendix 2 in section 3.3.3
- Clarification that the study kits will be created at Skanderborg Pharmacy (section 3.3.3 + 3.3.4)
- Clarification that the site investigator and the research nurse will also be responsible for study kits at each site (section 3.3.4)
- Change in exclusion criteria from "Extracorporeal circulation at the time of the cardiac arrest" to
   "Invasive mechanical circulatory support at the time of the cardiac arrest" (section 4.3)
- Minor change in the definition of hospital disposition (section 5.3)
- Addition of a reference to COSCA (section 5.3)
- Change in definition of vasopressor-free days (section 5.3)
- Addition of invasive ventilation-free days as a tertiary outcome (section 5.3)
- Change in the timepoints of SOFA score calculation from 4 and 24 hours to 24, 48, and 72 hours (section 5.3 + 7.2.4)
- Change in the definition of hyperglycemia (section 5.4.3)
- Change in definition of prior use of glucocorticoids from 5 days to 14 days (section 6.2.3)
- Addition of a subgroup analysis related to time from cardiac arrest to first study drug (section 6.2.3)
- Clarification that multiple imputation will only be performed if missing data is substantial (< 10%) (section 6.2.5)
- Clarification that data collection will not include the timing of the methylprednisolone dose (section 7.1)
- Removal of ethnicity as a variable (section 7.2.2)
- Removal of the reference to the updated IHCA Ustein guidelines (section 7.2.1)
- Addition of the Glasgow Outcome Scale Extended (section 7.2.4)
- Change in terminology from "legally authorized surrogate" and "next of kin" to "surrogate" (section 9.2.2 + 9.3.2)
- Clarification that the legal guardian cannot be related to trial procedures for the specific patient but can be involved in trial procedures for other unrelated patients (section 9.2.3 + 9.3.2)
- Update indicating approval by the regional ethics committee (section 9.3)

- Removal of sentence stating that data on non-enrollled patients can be obtained from DANARREST (section 11.3)
- Addition of Appendix 2
- Minor updates to Appendix 3
- Addition of Appendix 4
- Removal of Appendix 6 and 7
- Appendix 8 renumbered as Appendix 6 and updated

# Version 1.2 (Jan. 24, 2018) to 1.3 (Mar. 19, 2018)

- Change of the primary pharmacy to Skanderborg Pharmacy
- Addition details provided on the follow-up telephone interview (section 5.3)
- Clarification that the trial has been reported to the Danish Data Protection Agency (section 7.4)
- Clarification that consent after the cardiac arrest will be obtained by a physician (section 9.3.2)
- Addition of feasibility data from Odense (section 11.2)
- Clarification that shared data will be completely anonymized according to Danish law (section 13)

#### Version 1.1 (Jan. 24, 2018) to 1.2 (Jan. 24, 2018)

- Change of the primary pharmacy to Pharma Skan ApS
- Addition of Odense University Hospital as a site (multiple sections)

# Version 1.0 (Aug. 31, 2017) to 1.1 (Jan. 24, 2018)

- Corrections of minor typos and grammatical issues
- Clarification of the intervention being the combination of methylprednisolone and vasopressin (Overview, Trial flow chart)
- Clarification that the vasopressin placebo ampules and vasopressin ampules are identical (section 3.3.2)
- Production and labelling of the study kits at Pharma Skan ApS instead of the university pharmacy (section 3.3.3 and 3.3.4)
- Clarification that that the unblinded pharmacy staff will not be involved in outcome evaluation (section 3.4)
- Storage of medicine at room temperature as oppose to 2°C to 8°C (section 3.3.3)
- Clarification that the site investigator will keep track of study kits at each site (section 3.3.4)

- Clarification that data will also be obtained from the case report forms (section 3.5.1)
- Removal of E-Learning as a modality for education of study personnel (section 3.5.2)
- Clarification that patients who re-arrest in the emergency department can be included if they had sustained ROSC prior to the cardiac arrest (section 4.2)
- Definition of ROSC when patients are put on extracorporeal circulation redefined (section 5.1.1)
- Addition of the Glasgow Outcome Scale Extended for neurological outcome (section 5.3)
- Addition of a section of reporting of adverse events (section 5.4.6)
- Clarification of the follow-up after 90 days (section 5.5)
- Addition of a draft of the CONSORT flow diagram (section 6.2.1 + Appendix 3)
- Addition of two subgroup analyses according to the location of the cardiac arrest and the prior use of glucocorticoids (section 6.2.3)
- Addition of ordinal logistic regression (section 6.2.4)
- Various additions to the data collection (section 7.2)
- Clarification that the IDMC, the Good Clinical Practice unit, and regulatory agencies will have access to all relevant trial data (section 7.5)
- Clarification of the "legal guardian" (section 9)
- Clarification that consent for future data collection will be obtained from the legal guardian and the patient's next of kin if the patient is not able to provide consent (section 9.3.2)
- Clarification that the study results will be published irrespective of the results (section 12)
- Funding updates (overview and section 14)
- Removal of the section on potential expansion of the trial (section 15)
- Addition of Appendix 8: Charter for the independent data-monitoring committee (IDMC)

#### 1. BACKGROUND

# 1.1 In-hospital cardiac arrest

#### 1.1.1 Incidence and mortality

In-hospital cardiac arrest (IHCA) is relatively common with an estimated 200,000 treated cases in the United States each year.<sup>8</sup> Although no published data is currently available on the incidence of IHCA in Denmark, we estimate that approximately 2500-3000 IHCA occur each year. Unfortunately, outcomes remain poor with approximately 60% achieving return of spontaneous circulation (ROSC) and only 20-30% surviving to hospital discharge.<sup>9-11</sup> Furthermore, in initial survivors, there are substantial post-discharge morbidity and early mortality.<sup>10,12-14</sup>

# 1.1.2 An understudied entity

Clinical trials are sparse in cardiac arrest<sup>15,16</sup>, and especially in IHCA<sup>17</sup>, relative to the burden of the condition. In a systematic review of all randomized clinical trials involving cardiac arrest from 1995 to 2014, Sinha et al. found that 81 (88%) were exclusively in out of hospital cardiac arrest (OHCA), 7 (8%) involved OHCA and IHCA, and only 4 (4%) involved exclusively IHCA. The total number of included patients were 83 times higher in OHCA studies as compared to IHCA studies.<sup>18</sup>

Currently, there is a scarcity of evidence-based pharmacological interventions for IHCA.<sup>19-21</sup> The evidence for adrenaline (epinephrine) and amiodarone, the only two drugs currently recommended, is limited and based on extrapolation from OHCA.<sup>19-23</sup> There is therefore an, currently unmet, need for additional randomized clinical trials in IHCA in order to advance the science and improve patient outcomes.

# 1.1.3 Pathophysiology

In broad terms, cardiac arrest can be divided into three phases: pre-cardiac arrest, intra-cardiac arrest, and post-cardiac arrest, where intra-cardiac arrest can be further divided into a no-flow (no circulation) and a low-flow (circulation induced by chest compressions) phase. One of the main drivers of poor outcomes after cardiac arrest is the duration of the cardiac arrest (i.e. no-flow and low-flow time); for each minute increase in the length of the cardiac arrest, mortality substantially increases.<sup>24,25</sup> Because of this, and since ROSC is a prerequisite for more long-term survival, the main goal of intra-cardiac arrest interventions is to establish ROSC and limit the duration of the cardiac arrest.

The pathophysiology of cardiac arrest and the post-cardiac arrest syndrome is complex and has been described in extensive details elsewhere.<sup>26-28</sup> Ischemia during the cardiac arrest and subsequent ischemia-reperfusion injury activates multiple harmful pathways including systemic inflammation, endothelial

activation, activation of immunological and coagulation pathways, adrenal insufficiency, mitochondrial damage, and microvascular dysfunction.<sup>26</sup> Consequently this leads to a clinical state (the post-cardiac arrest syndrome) with global brain injury, impaired myocardial function, macrocirculatory failure, and increased susceptibility to infections.<sup>26</sup> Patient are often hemodynamically unstable following a cardiac arrest and early post-cardiac arrest hypotension is strongly associated with poor outcomes.<sup>29</sup>

# 1.2 Vasopressin

# 1.2.1 Pharmacology

Vasopressin (also known as antidiuretic hormone or arginine vasopressin) is a nonapeptide produced in the hypothalamus and secreted into the circulation through the posterior pituitary gland. Vasopressin exerts its effects through binding to one of its three receptor subtypes V1-V3. The V1 receptor mediates vasoconstriction, while binding to V2 mediates the antidiuretic effects in the kidney and activation of the V3 receptor in the pituitary gland stimulates the secretion of hormones. During states of shock, levels of vasopressin are low and exogenously administered vasopressin exerts profound vasoconstrictive effects. Where the vasoconstrictive effects of other vasopressors are reduced in conditions of hypoxia and acidosis the vasoconstrictive effects of vasopressin are maintained.<sup>30</sup> When administered intravenously, vasopressin has a half-life of approximately 10 to 35 minutes<sup>31,32</sup>

#### 1.2.2 Use outside cardiac arrest

Vasopressin is licensed in several countries, including the United States, Sweden, Germany, and the United Kingdom, to treat refractory shock in patient with sepsis. The 2016 Surviving Sepsis Guidelines recommends vasopressin as the second-line vasopressor after noradrenaline.<sup>33</sup> Vasopressin might also be beneficial in other forms of shock.<sup>34</sup> Terlipressin and desmopressin, synthetic vasopressin analogs with slower onset but longer duration<sup>35,36</sup>, are licensed in Denmark for the treatment of esophageal varices bleeding and diabetes insipidus, respectively.

#### 1.2.3 Use in cardiac arrest

The rationale for the use of vasopressin during cardiac arrest is based on studies demonstrating that plasma levels of vasopressin are lower in non-survivors compared to survivors<sup>37</sup>, and that vasopressin, through its potent vasoconstrictive properties, increases the coronary perfusion pressure and thereby the chance of ROSC.<sup>38,39</sup> These properties lead to clinical trials where vasopressin was compared to standard treatment.<sup>40-43</sup> Only one relatively small trial included IHCA patients.<sup>44</sup> In a meta-analysis of six randomized clinical trials,

there was no overall benefit of vasopressin administration during cardiac arrest.<sup>41</sup> However, there were a potential benefit in subgroups according to a first rhythm of asystole and early (< 20 minutes) drug administration.<sup>41</sup> In addition, a recent meta-analysis demonstrated that the administration of vasopressin increases the rate of ROSC and survival in patients with in-hospital arrest.<sup>43</sup> These latest findings are largely based on studies by Mentzelopoulos et al.<sup>45,46</sup> as described in more detail in section 1.4.

# 1.3 Methylprednisolone

# 1.3.1 Pharmacology

Methylprednisolone is a synthetic glucocorticoid which is a class of corticosteroids that is part of the larger group of steroid hormones. Glucocorticoids are produced in the adrenal cortex and exerts a wide range of functions in the body including regulation of metabolism, inflammation, and cell proliferation.<sup>47</sup> During situations with stress, glucocorticoids are secreted as a defense mechanism exerting widespread physiological functions.<sup>48</sup> The primary effect of glucocorticoids is exerted through binding to the glucocorticoid receptor followed by translocation to the nucleus where it modulates gene transcription through binding to glucocorticoid-responsive elements.<sup>49</sup> This is termed the genomic effects of glucocorticoids and it takes hours for a response to fully develop.<sup>50</sup> However, glucocorticoids also possess rapid (within minutes) non-genomic effects through interaction with cellular membranes and receptors, which are relevant in the setting of cardiac arrest.<sup>49-51</sup> Methylprednisolone is administered intravenously and has a biological half-life of approximately 12 to 36 hours.<sup>52</sup>

#### 1.3.2 Use outside cardiac arrest

Methylprednisolone is primarily licensed in Denmark as Solu-medrol® (Pfizer). Clinically, glucocorticoids have been used for decades in the treatment of various diseases due to its anti-inflammatory effects<sup>53</sup> and methylprednisolone is on the World Health Organization's list of essential medicines<sup>54</sup>. Glucocorticoids are used in several acute and critical conditions including bacterial meningitis, anaphylactic shock, and severe asthma or chronic obstructive pulmonary disease exacerbations. Glucocorticoids have been especially well-studied in the setting of septic shock where treatment with glucocorticoids increases shock reversal (i.e. weaning for vasopressor support) and may lower mortality.<sup>55</sup>

#### 1.3.3 Use in cardiac arrest

Studies in patients with cardiac arrest have demonstrated that levels of cortisol are higher in patients that are resuscitated when compared to patients that are not resuscitated which may illustrate an impaired

endocrine response in non-survivors. This is supported by animal studies where the administration of hydrocortisone during cardiac arrest increases ROSC rates.<sup>57</sup> This may relate to the cardiovascular effects of glucocorticoids which include increases in enzymes involved in adrenaline synthesis, inhibition of catecholamine re-uptake and breakdown, and by enhancement of cardiovascular sensitivity to catecholamines by increasing the binding capacity and affinity.<sup>48,58</sup> Data on glucocorticoid administration during human cardiac arrest is limited and small studies have shown conflicting results.<sup>59</sup>

# 1.4 The vasopressin, steroids, and epinephrine (VSE) trials

In two trials, published in 2009 and 2013, Mentzelopoulos et al. examined the effect of adding vasopressin and glucocorticoids to standard treatment in IHCA.  $^{45,46}$  In these two Greek, randomized, double-blind trials, the authors compared the addition of vasopressin (20 IU for each dose of adrenaline) and glucocorticoids (40 mg methylprednisolone) during cardiac arrest to placebo. After the cardiac arrest, patients in the intervention arm furthermore received glucocorticoids (300 mg hydrocortisone) if they had vasopressor-dependent shock. The results, which were published in the *Archives of Internal Medicine* (now *JAMA Internal Medicine*) and the *Journal of the American Medical Association (JAMA)*, were remarkable. The combined rate of ROSC was 148/178 (83%) in the intervention group vs. 118/190 (62%) in the control arm (p < 0.001). In the first trial, survival to hospital discharge was higher in the intervention group as compared to the placebo group (9/48 [19%] vs. 2/52 [4%], p = 0.02). In the second trial, the primary outcome of survival to hospital discharge with a favorable neurological outcome (cerebral performance category [CPC] score of 1 or 2) was higher in the intervention group as compared to the placebo group (18/130 [14%] vs. 7/138 [5%], p = 0.02). The authors also showed beneficial effects on post-cardiac arrest hemodynamics, organ failure, and inflammation.

#### 1.5 Guidelines regarding vasopressin and glucocorticoids

The VSE trials have received a great deal of attention in the literature with most commentaries arguing for external validation studies before clinical implementation. The International Liaison Committee on Resuscitation (ILCOR) reached the same conclusion: "Confidence in the treatment effects from bundled treatments [i.e. vasopressin and glucocorticoids] will increase if confirmed in further studies". The current American and European guidelines from 2015 do not recommend the routine use of vasopressin and glucocorticoids in IHCA primarily due to lack of trials externally validating the findings from the VSE trials. The American guidelines recognized the importance of this as a potential therapeutic option but specifically state "... further studies are needed before recommending the routine use of this therapeutic strategy".

#### 1.6 Standard of care

The standard of care during cardiac arrest is described by guidelines from the European Resuscitation Council and the American Heart Association. Pharmacological treatment is generally limited to amiodarone/lidocaine and adrenaline for patients with a refractory shockable rhythm and adrenaline for patients with a non-shockable rhythm. Although the evidence for amiodarone/lidocaine and adrenaline is limited and controversial these drugs are currently recommended and are given, when applicable, to most patients with cardiac arrest. The interventions of the current trial (vasopressin and methylprednisolone) will therefore be compared to placebo and both groups will receive the established standard of care consistent with the two VSE trials. 45,46

# 1.7 Post-cardiac arrest glucocorticoids

The intervention in the VSE trials included hydrocortisone for patients with vasopressor dependent shock 4 hours after the cardiac arrest. 300 mg of hydrocortisone was administered per day until shock reversal or for a maximum of 7 days. 45,46 For several reasons, this part of the intervention is not included in the current trial. First, considerable beneficial effects were seen in the original trials before the hydrocortisone was administered. This includes a substantial increase in ROSC as noted above, improvements in early hemodynamics, and an increase in 4-hour survival (intervention: 111/194 [57%] vs. placebo: 96/206 [47%], p = 0.01). 45,46 Second, a separate randomized clinical trial by members of our study team, not including the intra-cardiac arrest interventions, found no benefit of hydrocortisone for post-cardiac arrest patients with vasopressor dependent shock. 4 Third, assessing both intra- and post-cardiac arrest interventions combined does not allow for assessment of the individual effects of each intervention. If the current trial is positive, future trials are needed to then assess the post-cardiac arrest aspect of the VSE trials. Lastly, the primary outcome of the current trial is ROSC which will not be influenced by post-cardiac arrest treatment.

#### 2. TRIAL OBJECTIVES AND HYPOTHESES

<u>Primary objective</u>: To determine whether the combination of vasopressin and methylprednisolone, as compared to placebo, when administered during IHCA, will increase ROSC

<u>Hypothesis</u>: The combination of vasopressin and methylprednisolone administered during IHCA will increase ROSC

<u>Secondary objective</u>: To determine whether the combination of vasopressin and methylprednisolone, as compared to placebo, administered during IHCA will increase survival at 30 days and survival at 30 days with a favorable neurological outcome (CPC score 1 or 2)

<u>Hypothesis</u>: The combination of vasopressin and methylprednisolone administered during IHCA will increase survival at 30 days and survival at 30 days with a favorable neurological outcome (CPC score 1 or 2)

#### 3. TRIAL DESIGN

#### 3.1 Overview

This is an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, double-blind, superiority trial of vasopressin and methylprednisolone during adult IHCA. There will be 10 enrolling sites in Denmark. 492 adult patients with IHCA receiving at least one dose of adrenaline will be enrolled. The primary outcome is ROSC and key secondary outcomes include survival at 30 days and survival at 30 days with a favorable neurological outcome.

#### 3.2 Allocation

Patients will be randomized in a 1:1 ratio to either vasopressin and methylprednisolone or placebo in blocks with random sizes of 2, 4, or 6. The randomization will be stratified according to site.<sup>65</sup> An independent statistician will create the randomized allocation list using a random number generator. The list will only be shared with the pharmacy, which will not be involved in clinical care. The pharmacy and the independent statistician will both store the randomization list. As described in section 3.3 and section 3.4, sites will be provided with numbered blinded kits including either vasopressin and methylprednisolone or placebo ensuring allocation concealment.

#### 3.3 Interventions

# 3.3.1 Methylprednisolone and vasopressin

The study drugs will consist of 40 mg methylprednisolone (Solu-medrol®, Pfizer) and 20 IU of vasopressin (Empressin®, Amomed Pharma GmbH) given as soon as possible after the first dose of adrenaline. Additional doses of vasopressin (20 IU) will be administered after each adrenaline dose for a maximum of four doses (80 IU). The drugs will be produced, managed, and stored according to all relevant guidelines and regulations.

These drugs and doses are similar to the original VSE trial. However, for practical reasons (i.e. that one ampule of vasopressin contain two doses) this trial will include a maximum of four doses of vasopressin as compared to a maximum of five doses in the original trials. 45,46

#### 3.3.2 Placebo

The placebo for vasopressin will consist of 1 mL of 9 mg/mL NaCl ("normal saline") from 2 mL ampules identical to the vasopressin ampules. The placebo for methylprednisolone will also consist of 1 mL of 9

mg/mL NaCl. Normal saline is often administered to critically ill patients and have no effects or side-effects with these very small volumes.

#### 3.3.3 Procedures

The study drugs will be placed in a blinded study kit (a small box, see Appendix 2) containing one 40 mg dose of methylprednisolone (or placebo) and two 40 IU ampules (i.e. four 20 IU doses) of vasopressin (or placebo). The study kits will be prepared at Skanderborg Pharmacy, a company that specializes in the production of medicine and is approved by the Danish Health authorities, and shipped to the participating sites regularly. The study kit will be stored at room temperature and protected from light according to the manufacturers' instructions and brought to the IHCA by a designated member of the cardiac arrest team. Once it is anticipated that the patient will receive at least one dose of adrenaline, the kit will be opened, and the patient will be considered randomized. A designated member of the cardiac arrest team will then prepare the study drugs. Preparation of methylprednisolone will include mixing of the methylprednisolone powder (or placebo) with the solvent in a blinded manner (see section 3.4). The vasopressin (or placebo) will require no mixing. A visual guide showing the procedures will be placed in the kit and cardiac arrest team members will have training in the procedures (see section 3.5.2). We expect that these procedures will take approximately 1 minute and that they will not interfere with the clinical management of the patient. Once prepared, the drugs will be administered as soon as possible after the first dose of adrenaline; first the 20 IU (1 mL) vasopressin and then the 40 mg (1 mL) methylprednisolone (or their respective placebos). Additional doses of 20 IU vasopressin (or placebo) will be administered with each dose of adrenaline which is given every 3-5 minutes irrespective of the underlying rhythm.<sup>20</sup> A maximum of 4 doses of vasopressin (80 IU) will be administered. Only one dose of methylprednisolone will be administered.

# 3.3.4 Overview of study medication

Study kits will be produced and labelled centrally (Skanderborg Pharmacy). Study kits will be labelled with a unique ID consecutively according to site (e.g. 1XXX for site 1, 2XXX for site 2, etc.). The study kits and drugs will be clearly labelled according to standard practices for clinical trials (see Appendix 2). Study kits will be prepared and shipped to the participating sites on a regular basis. Once a study kit is opened, the site investigator, the research nurse, and the principal investigator will be informed. The central pharmacy will keep a tally of all study kits and make sure, along with the site investigator and the research nurse, that sites are always equipped with enough kits. The site investigator at each site will keep track of all delivered and used study kits. Data on actual drug administration (see section 3.3.3) will be entered in real-time on the

case report form and subsequently into the online database (see section 7). This will ensure optimal tracking of study drug delivery.

# 3.4 Blinding

The trial will be double-blind; patients, investigators, and the clinical team will be blinded to the allocation. Only the pharmacy providing the blinded, numbered kits will be aware of the allocation. The pharmacy will not be involved with clinical care or outcome evaluation.

Vasopressin placebo will consist of normal saline which, like vasopressin, is colorless and without any identifying features. The normal saline will be stored in 2 mL ampules that are identical to the vasopressin ampules. Furthermore, vasopressin has no distinctive rapid effects (except those related to the trial) resulting in possible identification. We therefore do not anticipate any risk of unblinding.

Methylprednisolone placebo will consist of an empty vial completely covered such that the clinical team cannot distinguish whether the vial is empty or contains the methylprednisolone powder. The methylprednisolone solvent or the NaCl placebo, which are identical in appearance, will be injected into the vial and the vial will be shaken to immediately dissolve the powder. The mixed solution will then be aspirated from the vial and administered to the patient. Since the mixed solution is colorless and without any identifying features, the clinical team will remain blinded to the treatment arm. A similar approach is being used in the ongoing SUP-ICU trial which is a multicenter, double-blind, randomized trial. <sup>66</sup>

In the blinded intervention kit, a sealed opaque envelope will contain the allocation assignment which will allow for emergency unblinding. The decision to unblind will be at the complete discretion of the treating physician and clinical team. However, we do not expect scenarios where emergency unblinding will be necessary. In case unblinding occurs, the reason(s) will be clearly documented in the case report form. The patient will remain in the trial.

# 3.5 Trial procedures

#### 3.5.1 Patients

The trial procedures will be limited to the interventions given during the cardiac arrest (see section 3.3) and the telephone interviews for long-term follow-up. (see section 5.3 and 5.5). There will be no planned blood draws, other interventions, or additional procedures. Data will be obtained from the study specific case report form, the electronic medical records, and the national Danish IHCA registry (DANARREST) (see section 7).

3.5.2 Clinical personnel

Prior to the beginning of patient enrollment and continuously throughout the enrollment period, the clinical

teams involved in IHCA resuscitation at the participating hospitals will be informed about the trial. Clinical

personnel will be informed about the background and objectives of the trial, the inclusion/exclusion criteria,

the interventions, and the trial procedures they are involved in (see section 3.3.3 and 9.3.2). A

demonstration of correct procedures using the study kits will be included. We anticipate formal, in-person

didactics quarterly with informal sessions and emails as applicable in between.

4. SETTING AND PATIENT POPULATION

4.1 Setting

The trial will be conducted at 10 hospitals in Denmark. All participating sites have clinical experience and

expertise in treating IHCA patients.

4.2 Inclusion criteria

Inclusion criteria:

1) IHCA

2) Age ≥ 18 years

3) Received at least one dose of adrenaline during CPR

Cardiac arrest is defined as unconsciousness, abnormal breathing, and a loss of pulses requiring chest

compressions and/or defibrillation. IHCA is defined as any individual with a cardiac arrest on hospital

grounds where the IHCA team is activated. This will include patients who re-arrest in the emergency

department or elsewhere after an OHCA if they, prior to the re-arrest, had sustained ROSC (i.e. spontaneous

circulation for at least 20 minutes).

These broad inclusion criteria were chosen to reflect the inclusion criteria in the two original VSE

trials. 45,46 The original trials included primarily patients with a non-shockable rhythm (84%). However, the

results were consistent and significant in both those with shockable and non-shockable initial rhythms and

there was no subgroup difference (p = 0.90, S. Mentzelopoulos, M.D., Ph.D., written communication, July

2017). We will therefore include IHCA patients with both shockable and non-shockable rhythms.

4.3 Exclusion criteria

Exclusion criteria:

- 1) Clearly documented "do-not-resuscitate" order prior to the cardiac arrest
- 2) Prior enrollment in the trial
- 3) Invasive mechanical circulatory support at the time of the cardiac arrest
- 4) Known or suspected pregnancy at the time of the cardiac arrest

Occasionally CPR is inadvertently started in patients with a pre-existing "do-not-resuscitate" order. If a "do-not-resuscitate" order is clearly documented in the electronical medical record prior to the cardiac arrest, the patient will be excluded. Patients previously included in the trial will be excluded to avoid statistical complexity related to correlated data. Since information on "do-not-resuscitate" orders and prior enrollment in the trial is documented (but might not be known by the cardiac arrest team) prior to the cardiac arrest and the intervention, any post-randomization exclusions will not lead to bias. <sup>67</sup> Mechanical circulatory support includes extracorporeal circulation and left ventricular assist devises. Patients having an IHCA while on mechanical circulatory support constitutes a very specific patient population with different characteristics and outcomes. They will therefore be excluded. Given that vasopressin and methylprednisolone are generally not recommended in pregnancy, patients with known or suspected pregnancy will be excluded. Cardiac arrest during pregnancy is exceedingly rare <sup>68</sup> and we expect that this exclusion criterion will lead to only few, if any, exclusions. If pregnant patients are included (i.e. if the pregnancy is not known and not obvious), we do not expect any harm to the patient or fetus. Guidelines recommend that cardiac arrest in pregnancy is treated according to usual guidelines including intra-cardiac arrest medications. <sup>69</sup>

#### 4.4 Co-enrollment

There will be no general restrictions on entry into other (post-cardiac arrest) clinical trials although this will be evaluated on a case-by-case basis.<sup>70</sup> We are not aware of any ongoing or planned trials in this patient population in Denmark.

#### 5. OUTCOMES

# 5.1 Primary outcome

#### 5.1.1 Definition

The primary outcome will be ROSC. ROSC will be defined as spontaneous circulation with no further need for chest compressions sustained for at least 20 minutes. This definition is consistent with the second VSE trial<sup>46</sup>, the *Get With the Guidelines® – Resuscitation* registry<sup>11</sup>, the Danish registry for IHCA (DANARREST)<sup>71</sup>, and the Utstein guidelines<sup>72</sup>. If a patient is placed on extracorporeal circulation during the cardiac arrest, the patient

will only be considered to have ROSC if they are able to be successfully weaned from the extracorporeal circulation with spontaneous circulation for at least 20 minutes.<sup>73</sup>

#### 5.1.2 Rationale

The rationale for any intra-cardiac arrest intervention is primarily to increase the rate of ROSC to subsequently improve the rate of meaningful survival. Since ROSC is a prerequisite for more long-term survival and since the focus of this investigation is intra-cardiac arrest interventions, ROSC is a logical and meaningful primary outcome. ROSC is a core outcome measure in both the IHCA<sup>72</sup> and OHCA<sup>73</sup> Utstein guidelines and is suggested as a potential primary outcome measure by the American Heart Association<sup>74</sup>.

# 5.2 Secondary outcomes

# 5.2.1 Definitions

The key secondary outcomes will be survival at 30 days and survival at 30 days with a favorable neurological outcome. A favorable neurological outcome will be defined as a CPC score of 1 or 2. The CPC score is a 5-point scale assessing neurological/functional outcomes after brain damage (Table 1).<sup>75</sup> Patients not alive at 30 days will be categorized as a poor neurological outcome.

| Table 1. Cerebral performance category (CPC) score | |
|---|---|
| Score | Definition |
| 1 | Good cerebral performance |
| - | Conscious, alert, able to work, might have mild neurologic or psychologic deficit. |
| | Moderate cerebral disability |
| 2 | Conscious, sufficient cerebral function for independent activities of daily life. Able to work in |
| | sheltered environment. |
| | Severe cerebral disability |
| 3 | Conscious, dependent on others for daily support because of impaired brain function. Ranges |
| | from ambulatory state to severe dementia or paralysis. |
| | Coma or vegetative state |
| 4 | Any degree of coma without the presence of all brain death criteria. Unawareness, even if |
| - | appears awake (vegetative state) without interaction with environment; may have |
| | spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness. |
| 5 | Brain death |
| , | Apnea, areflexia, electroencephalogram silence, etc. |

#### 5.2.2 Rationale

Survival at 30 days and survival at 30 days with a favorable neurological outcome are considered key outcome measures in cardiac arrest research.<sup>72-74</sup> The use of 30-day outcomes as compared to outcomes at hospital discharge avoids limitations related to potential difference in discharge practices.<sup>76-78</sup> The use of the CPC score is consistent with the second VSE trial<sup>46</sup>, the *Get With the Guidelines® – Resuscitation* registry<sup>11</sup>, and recommend by the Utstein guidelines<sup>72,73</sup> and the American Heart Association<sup>74</sup>.

# 5.3 Tertiary outcomes

Tertiary outcomes will include:

- 1) Vasopressor-free days
- 2) Invasive ventilation-free days
- 3) Sequential organ failure assessment (SOFA) score at 24, 48 and 72 hours
- 4) Hospital disposition
- 5) Modified Rankin scale (mRS) and Glasgow Outcome Scale Extended (GOSE) at 30 days
- 6) Health-related quality of life (EQ-5D-5L) at 30 days
- 7) 90-day outcomes:

Survival

Neurological outcome (CPC, mRS, GOSE)

Health-related quality of life (EQ-5D-5L)

The trial will include additional outcomes focused on hemodynamics, organ failure, additional measures of neurological outcome, and long-term outcomes.

To assess the potential beneficial effects of the intervention on hemodynamics, we will measure vasopressor-free days. A vasopressor will be defined as any continuous infusion of noradrenaline, dopamine, dobutamine, terlipressin, vasopressin, phenylephrine, and/or adrenaline. Vasopressor-free days will be defined as the number of days within the first 7 days after the cardiac arrest where the patient is not receiving vasopressors and is alive. Receiving vasopressors for at least 6 hours on a given day is defined as receiving vasopressors for that day. Contrary to other vasopressor outcomes, such as time to weaning from vasopressors, this outcome accounts for both vasopressor use and mortality. <sup>79</sup> Invasive ventilation-free days will be defined in a similar manner. Invasive ventilation is defined as mechanical ventilation through an endotracheal or tracheostomy tube.

To assess hemodynamics and organ failure, we will calculate SOFA score <sup>80</sup> at 24, 48 and 72 hours after the cardiac arrest in those alive. The SOFA score is a validated and widely used measure of organ failure assessing the respiratory, nervous, cardiovascular, hepatic, coagulation, and renal systems. <sup>80</sup> We will assess both the cardiovascular sub score as well as the overall SOFA score. The calculation of the SOFA score will be based on available clinical and laboratory data. Laboratory and clinical data closest to the given time point will be used. If a given component (e.g. bilirubin) is not available, it will be assumed to be within normal ranges. If PaO<sub>2</sub> values are not available, they will be imputed using imputations based on SpO<sub>2</sub> values. <sup>81,82</sup>

To further characterize neurological outcome and to allow for comparison with other trials and metaanalyses, the mRS<sup>83</sup> and GOSE<sup>84</sup> at 30 days and hospital disposition (e.g. home, rehabilitation, nursing home, hospice) will be collected. Hospital disposition will be defined at the time of discharge from the initial acute care hospital.

We will include 90-day survival as a measure of long-term survival. 90 days were chosen since it is unlikely that later mortality will be directly linked to the cardiac arrest or the trial interventions. 90 days is also consistent with recommendations from the American Heart Association.<sup>74</sup>

Both 30-day and 90-day survival will be obtained from the follow-up phone interview or the Danish Civil Personal Register which allows for accurate and virtually complete follow-up.<sup>85</sup> Neurological outcome (CPC, mRS and GOSE) and health-related quality of life (EQ-5D-5L<sup>86</sup>) at 30 and 90 days will be assessed via telephone communication with the patient or a surrogate. The telephone interview will be semi-structured and based on the GOSE and the EQ-5D-5L questionnaires. The interview will be conducted by a centrally located and trained member of the research team according to detailed standard operating procedures. In case the patient is still in the hospital, this interview will be face-to-face. In addition to CPC, both the mRS and health-related quality of life are recommended as outcome measures by the AHA.<sup>74</sup> Assessment of neurological outcome and health-related quality of life per telephone is valid and reliable.<sup>87,88</sup> A structured interview will be used to determine CPC, mRS, and GOSE.<sup>84</sup>

The mRS is a 7-point scale, ranging from 0 (no symptoms) to 6 (dead), assessing the degree of disability and dependence after a neurological injury such as stroke or cardiac arrest. A good outcome will be defined as a mRS of 0 to 3 and a poor outcome as 4 to 6. The GOSE is a 8-point scale that is an extension of the Glasgow Outcomes Scale (which is identical to the CPC, only with inverse scores) where the scores 1, 2 and 3 from the CPC score is divided into two.<sup>84</sup> The EQ-5D-5L is a well-established measure of health-related quality of life that is quantified as a utility (i.e. a measure of quality of life between 0 and 1). In addition to being a relevant outcome in itself, this will also allow for potential future cost-effectiveness analyses and comparison to the background population.

All outcomes recommended by the recent COSCA initiative (Core Outcome Set for Cardiac Arrest) are included in the current study.<sup>89</sup>

#### 5.4 Harm

#### 5.4.1 General consideration

Patients with IHCA have an in-hospital mortality of 70 to 80% and many patients experience post-cardiac arrest complications such as global brain injury, impaired myocardial function, macrocirculatory failure, and increased susceptibility to infections. <sup>26</sup> Furthermore, patients suffering from IHCA often have multiple underlying conditions including heart failure, myocardial infarction, respiratory insufficiency, diabetes, infections, and/or renal insufficiency. <sup>90</sup> The immediately preceding cause might be related to circulatory failure (e.g. cardiogenic shock, sepsis), respiratory failure (e.g. pneumonia, chronic obstructive pulmonary disease), arrhythmias (e.g. primary arrhythmias, myocardial infarction), or rarely neurological disorders. <sup>91-94</sup> Given this, it is difficult, if not impossible, to comprehensively report all adverse events and assess their possible relationship with the intervention in this patient population. Both vasopressin and methylprednisolone are considered safe and are commonly used in clinical practice. The overall benefit and potential harm of the interventions will be captured in our primary and secondary outcomes. Any specific adverse events suspected by the clinical team to be related to the intervention will be documented.

#### 5.4.2 Definitions

The following definitions will be used<sup>2</sup>:

<u>Adverse event</u>: any untoward medical occurrence in a subject to whom a medicinal product is administered and which does not necessarily have a causal relationship with this treatment

<u>Serious adverse event</u>: any untoward medical occurrence that at any dose requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital anomaly or birth defect, is life-threatening, or results in death

<u>Unexpected serious adverse reaction</u>: a serious adverse reaction, the nature, severity, or outcome of which is not consistent with the reference safety information

#### 5.4.3 Specific adverse events

To assess specific adverse and potentially serious adverse events (primarily related to methylprednisolone), we will collect data on the following:

- 1) Hyperglycemia (> 180 mg/dL or 10 mmol/L<sup>95</sup>) within the first 48 hours
- 2) Requirement for a continuous insulin infusion (≥ 1 hour) within the first 48 hours
- 3) Hypernatremia (> 145 mmol/L<sup>96</sup>) within the first 48 hours
- 4) New infections after the cardiac arrest during the hospital stay (defined below)
  - 4a) Bacteremia
  - 4b) Pneumonia
  - 4c) Urinary tract infections
- 5) New or changing antibiotics after the IHCA during the hospital stay
- 6) Clinical diagnosis of gastrointestinal bleeding after the IHCA requiring at least one blood transfusion during the hospital stay
- 7) Acute mesenteric ischemia based on a clinical diagnosis (signs and symptoms, colonoscopy and/or radiology findings) leading to surgery<sup>97</sup>
- 8) Peripheral (i.e., limps or digits) ischemia based on a clinical diagnosis (signs and symptoms and/or radiology findings) leading to surgery

Assessment of adverse events will be based on available laboratory values and clinical data. No specific procedures or blood draws will be performed.

Given the complexity of the post-cardiac arrest syndrome, it is difficult to diagnose and precisely define new infections in this patient population. For example, the new Sepsis-3 definitions<sup>98-100</sup> do not readably apply since many post-cardiac arrest patients will have a change in SOFA score  $\geq 2$  irrespective of any ongoing infection. Furthermore, fever is difficult to assess during the early post-cardiac arrest period where targeted temperature management is often utilized. Infections included here are therefore restricted to those that can be, at least partly, objectively defined and those that are the most common after cardiac arrest. <sup>101,102</sup> Bacteremia will be defined as a positive blood culture (not including presumed contamination or non-pathogenic bacteria not leading to antibiotics) obtained after the cardiac arrest. Pneumonia will be defined as new or progressive consolidation on a chest radiograph and at least two of the following: fever (>  $38^{\circ}$ C), leukocytosis (white blood cell count  $\geq 12,000$  cells/µL) or leukopenia (white blood cell count < 4,000 cells/µL), or the presence of purulent tracheobronchial secretions. <sup>103,104</sup> Urinary tract infection will be

defined as a positive urine culture (≥ 100,000 colony-forming units/mL from a pathogenic organism) obtained after the cardiac arrest.<sup>105</sup>

#### 5.4.4 Timeline

Vasopressin has a half-life of approximately 10 to 35 minutes<sup>31</sup> and methylprednisolone has a biological half-life of approximately 12 to 36 hours<sup>52</sup>. There is therefore no anticipation of adverse events after hospital discharge as patients with IHCA have long hospital stays.<sup>106</sup> The above mentioned adverse events will therefore only be assessed during the hospital stay.

#### 5.4.5 Suspected Unexpected Serious Adverse Reaction (SUSAR)

Suspected Unexpected Serious Adverse Reactions (SUSAR) will be reported to the independent data-monitoring committee (IDMC) (see section 10.2) and the regulatory authorities as applicable. Given the consideration outlined in section 5.4.1, most events or conditions, including but not limited to organ failure, infection, tissue ischemia, brain damage, cardiac arrest, and death, will not be considered SUSARs. This approach is compatible with an ongoing international, multicenter trial in post-cardiac arrest (ClinicalTrials.gov Identifier: NCT02908308). No events, including those outlined in section 5.4.3, will automatically lead to unblinding.

# 5.4.6 Reporting

Once a year the sponsor will submit a list of all registered adverse events that have occurred during the trial period as a well as a report on safety of the trial subjects to the Danish Medicines Agency. The sponsor will notify the Danish Medicines Agency when the trial has been completed (no later than 90 days thereafter) or if earlier than planned, the reasons for stopping the trial must be given. The results from the clinical trial including important adverse events will be recorded on EudraCT.

# 5.5 Additional follow-up

The primary trial and publication will be related to the study outcomes (section 5.1, 5.2, and 5.3). However, extended follow-up at six months and 1 year, including overall survival, neurological outcomes, and health-related quality of life, will be collected and reported. Data will be collected and analyzed like the 90-day outcomes and will be reported in a separate publication. Although the overall trial will be unblinded after the collection of the 90-day outcomes, the person assessing six months and 1-year outcomes will be blinded to treatment assignment.

#### 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN

#### 6.1 Sample size calculation

The trial will be powered to the primary outcome of ROSC. In the original trials, the combined rate of ROSC was 148/178 (83% [95%CI: 77%, 88%]) in the intervention group and 118/190 (62% [95%CI: 55%, 69%]) in the placebo group for an absolute risk difference of 21% and a relative risk of 1.34. <sup>45,46</sup> For this trial, we assume a ROSC rate of 45% in the control group (based on preliminary data from some of the participating sites [see section 11.2]). We assume an absolute difference of 13% between the control and intervention group corresponding to a ROSC rate of 58% in the intervention group and a relative risk of 1.29. With these estimates, an alpha of 0.05, and the use of the chi-squared test, we will need a total of 492 patients (i.e. 246 in each group) to have 80% power to detect a statistically significant difference between groups.

With an estimated survival rate of 20% (see section 11.2), an alpha of 0.05, and the use of the chi-squared test, the power of the trial to detect a significant difference between groups is illustrated in Figure 1 according to various estimates of treatment effect (i.e. risk ratios). Of note, the risk ratio for survival to hospital discharge was 4.87 (95%CI: 1.11, 21.4) in the first VSE trial and 2.73 (95%CI: 1.18, 6.32) for survival to hospital discharge with a favorable neurological outcome in the second VSE trial. 45,46 The trial will have  $\geq$  98% power to detect a risk ratio of  $\geq$  1.80 with a survival rate of 20% or higher in the placebo group. Sample size and power was calculated with PROC POWER in SAS v. 9.4 (SAS Institute, Cary, NC, USA).



Figure 1. Relationship between treatment effect (risk ratio) for survival and trial power
#### 6.2 Statistical analysis plan

#### 6.2.1 General considerations

The statistical analyses and reporting will adhere to the CONSORT guidelines. All tests will be two-sided, a P value < 0.05 will be considered significant, and all confidence intervals will have 95% coverage. P values will only be reported for the primary outcome and the two key secondary outcomes.

Patient inclusion and exclusion will be illustrated in a CONSORT flow diagram (see Appendix 3 for a draft). All analyses will be conducted on a modified intention-to-treat basis only including patients receiving the

pregnancy). In a double-blind trial, this approach is unbiased while increasing precision. <sup>67</sup>

The two groups will be compared in relation to baseline patient and cardiac arrest characteristics using descriptive statistics.

first dose of the study drug and meeting all inclusion criteria and no exclusion criteria (except criteria #4:

The persons conducting the statistical analysis will be blinded to the randomized allocation and the statistical analysis will be performed separately by two investigators. Groups will be designated as "A" and "B" until all pre-specified analyses are performed and shared with all authors and the IDMC (see section 10.2).

## 6.2.2 Primary and secondary outcomes

The primary and secondary outcomes (binary variables) will be presented as counts and proportions in each group. Results will be reported as both risk ratios and risk differences. 95% confidence intervals will be obtained using methods described by Miettinen and Nurmimen. <sup>109</sup> In case results are significantly different between groups, the number needed to treat (with 95% confidence intervals) will also be provided. P values will be obtained from Fisher's Exact test.

As a sensitivity analysis, we will estimate the risk ratio with 95% confidence intervals for the primary outcome while adjusting for center and strong prognostic factors, specifically age, whether the cardiac arrest was witnessed, and the initial rhythm, as covariates. 110-113 Small centers (i.e. those with less than 30 patients included) will be combined. The risk ratio will be estimated from a log-binomial regression model. 114 If this model fails to converge, a modified Poisson regression model will be used instead. 114,115 Age will be included as a linear continuous variable and the initial rhythm as a binary variable (shockable or non-shockable).

#### 6.2.3 Subgroup analyses

Subgroup analyses will be performed on both the absolute and relative scale. The analyses will include five pre-defined subgroup analyses for the primary and key secondary outcomes according to 1) first

documented rhythm, 2) whether the cardiac arrest was witnessed, 3) patient age (dichotomized by the median), 4) time from cardiac arrest to first study drug (dichotomized by the median), and 5) time from adrenaline administration to first study drug (dichotomized by the median). First documented rhythm will be categorized as non-shockable (i.e. asystole or pulseless electrical activity) or shockable (i.e. ventricular fibrillation or pulseless ventricular tachycardia). The trial is not powered to detect subgroup differences, and these will be considered exploratory and hypothesis generating.

#### 6.2.4 Addition analyses and outcomes

For the tertiary outcomes vasopressor-free days, SOFA scores, and health-related quality of life (continuous variables) differences between groups will be estimated using a linear regression model. SOFA scores and health-related quality of life will only be assessed in those alive at the time of measurement.

Survival until 90 days will be presented with Kaplan-Meier curves but will otherwise be analyzed as a binary outcome as described in section 6.2.2

Adverse events and other binary outcomes will be presented and analyzed like the primary and secondary outcomes.

As additional exploratory analyses, ordinal neurological outcomes (i.e. CPC, mRS, GOSE) will be analyzed using ordinal logistical regression. <sup>124</sup> Before these analyses, the proportional odds assumption will be tested. In case the proportional odds assumption is not met, ordinal logistical regression will not be performed, and data will be presented descriptively.

#### 6.2.5 Missing data

Missing data will be reported in the relevant publications. We do not expect any missing data for the primary outcome or the key secondary outcomes. For mortality up to 90 days, there may be some very limited loss to follow-up. We do not expect missing data on the vasopressor-free days, SOFA scores, or adverse events. There might be some limited missing data for neurological outcomes and health-related quality of life at 90 days (and potentially at 30 days) due to loss to follow-up. Multiple imputation using known risk factors for outcomes after IHCA will be used to impute values for patients with missing data if missing data is substantial (> 10%).

## 6.2.6 Multiple comparisons

No adjustments will be made for multiple comparisons. The rationale for this approach is three-fold. First, the trial has a clearly defined primary outcome which will ensure that the risk of a Type I error (i.e. false positives) is equal to the set alpha (i.e. 0.05) for this outcome. Second, the simplest procedure to control the

family-wise error rate is the Bonferroni correction where the alpha is divided by the number of tests performed within the "family" of tests. However, defining the "family" is difficult and at best arbitrary. Third, any adjustment for multiple comparisons to control the family-wise error rate increases the chance of Type II errors (i.e. false negatives). Given that the risk of Type I errors is not well defined when conducting multiple secondary analyses, these specific analyses should be considered exploratory and hypothesis generating.

#### 6.2.7 Statistical stopping criteria

Since the primary outcome is not mortality, there will be no formal stopping criteria for efficacy. There will be no predefined stopping criteria for futility since enrollment of the full cohort might allow for detection of efficacy in subgroups or in other outcomes even if the primary outcome is neutral. Furthermore, since two previous randomized clinical trials have shown efficacy<sup>45,46</sup>, a neutral trial with an adequate sample size will be important. For potential stopping due to safety concerns, see section 10.2.

#### 7. DATA COLLECTION AND MANAGEMENT

## 7.1 Data collection process

A trained research nurse, along with the site investigators, will be responsible for data collection and entry. Very limited data will be obtained from the clinical cardiac arrest team in real-time on a numbered case report form (see Appendix 4) that accompanies the study kit. This will include the patient identifier (i.e. CPR number), timing of the first adrenaline dose, timing of the first vasopressin dose, and the total doses of vasopressin administered. This, along with the telephone interviews for long-term follow-up, will be the only source data and all additional data will be obtained from the electronical medical records or DANARREST (see section 7.6) and will be based on measurements and assessments made by the clinical team. Data will be entered directly into the database software (see section 7.4).

## 7.2 Variables

## 7.2.1 Overview

All IHCA patients at the participating sites will be entered into a screening log. For those not randomized, a specific reason for non-inclusion/exclusion will be documented. All randomized patients who received the study drug will be entered into the main database.

A detailed data dictionary that clearly defines all included variables will be created prior to patient enrollment. The data dictionary will provide the name of the variable (including the code used in the

database), a detailed definition of the variable, categories for categorical variables, and units and ranges for continuous variables.

The number of collected variables will be kept relatively small to limit resource use and data entry mistakes. The included variables largely follow the IHCA Utstein guidelines from 1997.<sup>72</sup> Below is provided a brief overview of the included variables but details are reserved for the data dictionary.

## 7.2.2 Pre-cardiac arrest characteristics

Trial related variables

Study ID

Site

Receipt of study medication

If no, reason for no study medication provided

Doses of study medication provided

Requirement for emergency unblinding

Inclusion criteria

**Exclusion criteria** 

Date and time consent for data collection is obtained

## Patient demographics and characteristics

Name

Unique patient identifier (CPR number)

Age

Sex

Race

Height

Weight

# Conditions/medications prior to the cardiac arrest

Co-morbidities (cardiac and non-cardiac)

CPC score and mRS prior to current hospital admission

Reason for admission

Length of stay prior to the cardiac arrest

Receipt of glucocorticoids within the last month

Use of oral or intravenous glucocorticoids during the current admission Previous IHCA during this admission

#### 7.2.3 Cardiac arrest characteristics

Location and time

Location of the cardiac arrest

Date and time of the cardiac arrest

# Interventions in place

Vasopressors

Mechanical ventilation

Intravenous access

Renal replacement therapy

# Cardiac arrest variables prior to the intervention

Presumed cause of the cardiac arrest

Initial rhythm

Witnessed

Time to first rhythm analysis

## Cardiac arrest variables after the intervention

Date and time of the end of resuscitation (ROSC or termination without ROSC)

# 7.2.3 Post-cardiac arrest characteristics

Targeted temperature management

If yes, target temperature and duration

Cardiac catheterization, percutaneous coronary intervention, and coronary artery bypass grafting

Procedures related to neurological prognostication (e.g. EEG, imaging, biomarkers)

Use of intravenous glucocorticoids

Renal replacement therapy

Adverse events (see section 5.4.3)

7.2.4 Outcomes

**ROSC** 

SOFA scores at 24, 48, and 72 hours

Vasopressor-free days

Hospital disposition

Survival at 30 and 90 days

CPC score at 30 and 90 days

mRS at 30 and 90 days

Glasgow Outcome Scale Extended at 30 and 90 days

EQ-5D-5L at 30 and 90 days

# 7.3 Data quality and validity

Data quality and validity will be optimized by having a single trained research nurses enter all data according to a detailed data dictionary. REDCap (see section 7.4) is designed such that data forms contain field-specific validation checks ensuring that mandatory fields are filled out and that continuous variables are within predefined ranges. Given its limited utility, double-data entry will not be performed.<sup>127,128</sup>

#### 7.4 Data storage and security

The database application we will use is REDCap.<sup>129</sup> REDCap is a professional database that provides a user-friendly interface. The REDCap data management system is secure, fully compliant with all regulatory guidelines, and includes a complete audit-trail for data entry validation. Through these mechanisms, as well as relevant training for all involved parties, patient confidentiality will be safeguarded. REDCap is available for free at participating sites.

The short paper case report form and the consent form for each patient will initially be stored in a secure, locked place at the individual sites. Every half year these will be transported to the Research Center for Emergency Medicine in Aarhus while a copy will remain at the sites. Here they will be securely stored in locked cabinets, where only the principal investigator and the research nurse will have access. The files will be stored for 5 years after the end of the trial, where after they will be destroyed.

The trial has been reported to the Danish Data Protection Agency.

#### 7.5 Data access

During the trial, the principal investigator and the research nurse will have access to the entire database, while site investigators will have access to data from their own sites. Once the database is locked, a deidentified version of the database will be made available to the members of the steering committee. The IDMC, the Good Clinical Practice unit, regulatory agencies, and other relevant entities will have direct access to patients' records and to all relevant trial data including the case report form as applicable.

#### 7.6 DANARREST

For the intra-cardiac arrest characteristics, data is captured in real-time by the clinical cardiac arrest team as part of a nationwide quality improvement registry (DANARREST).<sup>9,71</sup> DANARREST is a quality improvement registry that aims to track the epidemiology of IHCA in Denmark. All hospitals in Denmark will participate within a few years and the clinical personnel are required to enter data. A Danish version of the DANARREST case report form is provided in Appendix 5.

#### 8. CLINICAL TREATMENT

The clinical management of included patients will be at the complete discretion of the treating clinical team in order to test the interventions in a real-life clinical scenario. In general, management will adhere to the intra- and post-cardiac arrest guidelines provided by the European Resuscitation Council<sup>130</sup> and the Danish Resuscitation Council<sup>131</sup> but no specific treatments will be prohibited or mandated. The sites will be informed about the most recent guidelines for intra-cardiac arrest care and will be encouraged to limit premature termination of resuscitation efforts.<sup>132</sup> Sites will also be encouraged to follow European Resuscitation Council post-cardiac arrest guidelines<sup>95</sup> including appropriate neurological prognostication.

# 9. ETHICAL CONSIDERATIONS

## 9.1 Clinical equipoise

#### 9.1.1 Potential benefits

Details about the potential benefits of the intervention are provided in the background section (section 1.2, 1.3, and 1.4). In brief, randomized controlled trials, primarily in the OHCA setting, have found no benefit or harm of sole vasopressin administration.<sup>41</sup> The data on steroid administration during cardiac arrest is more limited and have shown conflicting results although no study has shown harm.<sup>59</sup> The combination of

vasopressin and glucocorticoids has been tested in two randomized, double-blind trials finding significant and meaningful increases in ROSC, survival, and survival with a favorable neurological outcome. 45,46

#### 9.1.2 Potential harms

The two VSE trials found no signs of significant harm with the combination of vasopressin and glucocorticoids during cardiac arrest. <sup>45,46</sup> In the first VSE trial there was an increase in the number of hyperglycemic episodes on day 2 and 3 in the intervention arm. <sup>45</sup> In the second VSE trial, there was a small increase in the proportion of patients receiving post-cardiac arrest insulin in the intervention arm. <sup>46</sup> Randomized clinical trials in other intensive care unit populations such as those with sepsis have found a small increase in hyperglycemia and hypernatremia, but no increased risk of infections, gastrointestinal bleeding, or muscular weakness, with small to moderate doses of glucocorticoids. <sup>55,133,134</sup> The idea that glucocorticoids could impair cardiac healing after myocardial infarction is based on old case reports. <sup>135</sup> A meta-analysis of controlled trials of glucocorticoids in patients with acute myocardial infarction found no association with myocardial rupture and in fact noticed a decrease in mortality with the administration of glucocorticoids. <sup>136</sup>

## 9.1.3 Risk/benefit ratio

From the data provided above in section 9.1.1. and 9.1.2 and in the background section (section 1.2, 1.3, and 1.4), the current risk/benefit ratio is encouraging for vasopressin and methylprednisolone administered during IHCA. However, given the potential lack of generalizability of the two VSE trials, international guidelines are currently not recommending this treatment but instead calls for additional clinical trials. <sup>19-21</sup> Taken together, there is clear clinical equipoise for the combination of vasopressin and methylprednisolone during IHCA.

#### 9.2 Research in cardiac arrest

#### 9.2.1 General considerations

Research in cardiac arrest is ethically challenging for two reasons: 1) Patients are unconsciousness and can therefore not provide informed consent and 2) treatment must be administered within minutes limiting the possibility of obtaining informed consent from a legally authorized representative. <sup>137,138</sup> Despite these challenges, there is an ongoing need to conduct research in this, and similar, patient populations to improve outcomes. International guidelines, such as the revised Declaration of Helsinki<sup>1</sup>, European regulations<sup>2</sup>, and

the Good Clinical Practice guidelines<sup>3</sup>, clearly supports research in such populations. For example, the revised Declaration of Helsinki states:

"Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorised representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorised representative."

The current trial will adhere to the revised Declaration of Helsinki as well as all applicable laws and regulatory guidelines.

## 9.2.2 Danish regulations

Danish law allows research without informed consent in situation where the following criteria are met<sup>139,140</sup>:

- 1) The research can only be conducted in the given acute situation
- 2) The patient is incapable of providing informed consent
- 3) Consent cannot be obtained from a surrogate given the urgency of the intervention
- 4) The research specifically involves the patient's current condition
- 5) There is a possibility of benefit to the patient

The current trial fulfils all the above criteria as described in section 9.2.3 for #1-4 and for #5 in section 9.1. Under these circumstances, research with pharmacological interventions is allowed if the following is obtained 139-141:

- 1) Consent is obtained from a designated "legal guardian" ("forsøgsværge" in Danish)
- 2) Informed consent is obtained from the patient or a surrogate as soon as feasible

A "legal guardian" is a physician not involved in the research related to the specific patient and who are not in an inferior/superior position to the investigator/sponsor, who should act according to the interest of the research participant.

## 9.2.3 Regulations in relation to the current trial

#1. The research can only be conducted in the given acute situation

Given the high morbidity and mortality of IHCA (see section 1.1.1), clinical trials are highly needed to improve patient outcomes. Animal studies do not adequately reflect the clinical condition of cardiac arrest and human trials are needed to advance the treatment of cardiac arrest patients. There is no other clinical condition that reflects cardiac arrest and any study aimed to improve outcomes for cardiac arrest patients can therefore only be conducted in this population.

#2. The patient is incapable of providing informed consent

IHCA is an unpredictable and sudden event that often occurs in patients that are already acutely sick. It is therefore impossible to obtain consent prior to the event. During the cardiac arrest, patients are unconscious and therefore not able to provide consent.

#3. Consent cannot be obtained from a surrogate given the urgency of the intervention

Cardiac arrest is an acute event that often lasts for less than 30 minutes. The intervention will be administered as soon as possible after the first adrenaline dose, which is given as soon as possible in patients with a non-shockable rhythm (most often < 5 minutes from the beginning of the cardiac arrest 143) and after the third defibrillation in patients with a shockable rhythm (approximately 6-7 minutes after the beginning of the cardiac arrest 20). Given these time frames, it would be impossible to obtain consent from a surrogate.

#4. The research specifically involves the patient's current condition

The interventions in this trial is specifically targeted for IHCA patients and if proven effective, will benefit this patient population.

#### 9.3 Procedures

9.3.1 Ethical review committee

The trial has been approved by the regional ethics committee (case number: 1-10-72-42-18).

## 9.3.2 Trial-specific procedures

The "legal guardian" will be either a physician member of the cardiac arrest team or a physician on call and available 24/7. The physician might be involved in the clinical care of the patient but will not be involved in trial procedures related to the specific patient. The legal guardian can be involved in trial procedures for other unrelated patients. Through ongoing training and information (see section 3.5.2), the "legal guardian" will be aware of the trial including the background and significance, inclusion/exclusion criteria, and potential risks and benefits. This way, the "legal guardian" will be able to make an informed and prompt decision about patient enrollment. The specific details related to the "legal guardian" (i.e. who will be the designated "legal guardian") will be site-specific.

As soon as possible, consent for future data collection will be obtained by a physician from the patient or if the patient is not able to provide consent, then by the legal guardian and a surrogate. The consent form will be signed by the patient or a surrogate and the person obtaining the consent. If a patient dies before it is possible to obtain consent (we anticipate that approximately 50% will not survive the cardiac arrest, see section 6.1), patient data will be included in the trial. If a patient denies future participation in the trial, no additional data will be collected but all data collected up until the point of withdrawal will be included consistent with Danish law.

When approached, the patient or a surrogate will be informed, verbally and in writing, about the background and significance of the study, inclusion criteria, potential risks and benefits, as well as a brief description of the study protocol. They will be informed that no additional interventions or procedures, except the telephone interviews for long-term follow-up, will be performed and that future participation will only include data collection. The patient or the surrogate will then provide written informed consent utilizing the informed consent form approved by the ethical review committee. When consent is obtained from participants or a surrogate, information about potential de-identified data sharing will also be included.

#### 9.3.3 Insurance

The patients in the study are covered by the Danish patient insurance. 146

#### **10. MONITORING**

## 10.1 Good Clinical Practice monitoring

The sites will be monitored by the regional Good Clinical Practice monitoring units affiliated with the participating sites. A detailed monitoring plan will be developed prior to trial commencement.

## 10.2 Independent data-monitoring committee (IDMC)

The IDMC will be responsible for safeguarding the interests of trial participants, assessing the safety and efficacy of the interventions during the trial, and for monitoring the overall conduct of the clinical trial. The IDMC will consist of three individuals: two clinicians/trialist with expertise in cardiac arrest/critical care research and a biostatistician/epidemiologist. The IDMC members will be chosen such to avoid any financial or intellectual conflicts of interest. The IDMC will be independent from the sponsor and the trial investigators. The IDMC will review deidentified data on a yearly basis (or more often if determined by the IDMC) for safety; unless there are group differences necessitating unblinding (as determined by the IDMC), the IDMC will be blinded to treatment groups. The trial will continue while the IDMC review data. After the yearly review, the IDMC will create a short report to the steering committee with recommendations for continuation, modifications, or termination of the trial. As noted in section 6.2.7, there will be no formal stopping criteria for efficacy or futility. Criteria for recommending termination will be at the discretion of the IDMC and there will be no formal statistical criteria for termination due to safety. The final decision regarding potential modifications or termination will rest with the steering committee and the principal investigator. A detailed charter for the IDMC is provided in Appendix 6.

## 11. TIMELINE AND ENROLLMENT

## 11.1 Timeline



## 11.2 Feasibility

Data from 2016 from five of the participating hospitals are provided in Table 2. As illustrated, we expect that approximately 457 patients will be eligible for enrollment each year. Given the acuity of IHCA, we do not assume that all eligible patients will be enrolled. However, given the large number of eligible patients, we will reach our target sample size over approximately 3 years of active enrollment (see section 11.1) with an enrollment rate as low as 35%. With the addition of more sites, we expect enrollment to happen faster.

| | IHCA with | IHCA with ≥ 1 dose of | ROSC in IHCA | 30-day survival in |
|---|---|---|---|---|
| Hospital | indication for | adrenaline given (i.e. | with ≥ 1 dose of | IHCA with ≥ 1 dose |
| | CPR | target population) | adrenaline given | of adrenaline given |
| Aarhus – Skejby* | 100 | 58 | 21 (36%) | 11 (19%) |
| Randers | 75 | 56 | 16 (29%) | 7 (13%) |
| Aalborg – South | 208 | 132 | 60 (45%) | 22 (17%) |
| Rigshospitalet | 198 | 177 | 80 (45%) | 33 (19%)** |
| Odense | 63 | 34 | 15 (44%) | 8 (24%) |
| Total | 644 | 457 | 192 (42%) | 81 (18%) |

<sup>\*</sup> This site is currently expanding as it is merging with two other hospitals. We therefore expect a higher number of annual IHCA at this site.

#### 11.3 Enrollment

Enrollment at each site will be continuously monitored by the site investigator, the research nurse, and the principal investigator. Formal reports outlining the number of IHCA and the proportion of those enrolled at each site will be shared with the steering committee quarterly. In case multiple eligible IHCA are not enrolled, a root cause analysis will be performed, and efforts will be made to avoid such issues in the future. Given the urgency of IHCA, we do not expect 100% enrollment of eligible IHCA. However, we will aim for enrollment of > 50% of eligible IHCA. In case that a site continuously underperforms despite troubleshooting and feedback, the steering committee will evaluate whether enrollment will continue at that site.

<sup>\*\*</sup> Estimated based on the ROSC rate and data from the other sites

#### 11.4 Additional sites

In case target enrollments are not met after 6 months to 1 year of enrollment, additional sites, in Denmark or outside Denmark, will be included. The principal investigator and the steering committee have multiple national and international ongoing collaborations allowing for recruitment of new sites.

#### 12. PUBLICATION PLAN

Three manuscripts are planned from the current trial. Prior to unblinding of the results, a methodology article will be published including a detailed description of the trial and the statistical analysis plan. The second and primary manuscript will include the main results including pre-defined primary, secondary, and tertiary outcomes. The manuscript will adhere to the CONSORT guidelines. The principal investigator will be the first and corresponding author. Additional authorship will follow authorship guidelines from the International Committee of Medical Journal Editors and will include members of the steering committee. In addition, as a guideline, sites enrolling > 50 patients will be entitled one additional author and sites enrolling > 100 patients two additional authors in addition to the site investigators and members of the steering committee. The trial results will be shared with participating sites and via press releases but not directly with the participating patients. The third manuscript will include long-term follow-up at six months and 1 year (see section 5.5). Study findings will be published irrespective of the results.

#### 13. DATA SHARING

Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. Data will be completely anonymized according to Danish law.

All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing. Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors<sup>147</sup> and might or might not include authors from the steering committee depending on the nature of their involvement.

14. FUNDING

Funding for the trial is provided by Aarhus University Research Foundation (kr. 3,000,000), the Department

of Clinical Medicine, Aarhus University (kr. 950,000), the Central Denmark Region (kr. 55,751), and the

Independent Research Fund Denmark (kr. 2,343,495). Empressin® and corresponding placebo ampules are

provided free of charge by Amomed Pharma GmbH. The funding agencies and Amomed Pharma GmbH have

no role in the design and conduct of the study; collection, management, analysis, and interpretation of the

data; preparation, review, or approval of the manuscript; or the decision to submit the manuscript for

publication.

**15. TASKS AND RESPONSIBILITIES** 

Principal investigator and sponsor: Overall responsibility for protocol development, funding, budget

overview, data dictionary development, ethical approval, trial registration, daily management, trial

oversight, contact to the pharmacy, contact to Good Clinical Practice monitoring unit and the data and safety

monitoring board, assessment of overall recruitments, potential recruitment of additional sites, data

analysis, and dissemination and presentation of results

Steering committee: Protocol development, funding, budget overview, data dictionary development, trial

oversight, dissemination of results, responsibilities as principal investigator for short time periods

Site investigators: Responsible for site-specific enrollment, evaluation of eligible patients not included,

education of personnel at participating sites, reporting of site-specific issues or challenges to the principal

investigator, participant consent for data collection

Research nurse: Daily management, education of personnel at participating sites, contact to pharmacy,

contact to Good Clinical Practice monitoring unit, data dictionary development, trial registration, data entry

and management, patient follow-up, budget overview

Clinical team: Administration of the study drug, participant consent for data collection

Good Clinical Practice-unit: See section 10.1.

Data and safety monitoring board: See section 10.2.

#### References

- World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. *JAMA*. 2013;310(20):2191-2194.
- The European Parliament and the Council of the European Unit. Clinical Trials Regulation (CTR) EU
   No 536/2014. 2014; https://ec.europa.eu/health/sites/health/files/files/eudralex/vol-1/reg\_2014\_536/reg\_2014\_536\_en.pdf. Accessed July 18, 2017.
- 3. ICH Harmonised Tripartite Guideline. Integrated Addendum To ICH E6(R1): Guideline For Good Clinical Practice E6(R2). 2016; http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E6/E6\_R2\_\_Step 4.pdf. Accessed June 30, 2017.
- 4. ICH Harmonised Tripartite Guideline. General Considerations for Clinical Trials E8. 1997; http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E8/Step4/E8\_Guideline.pdf. Accessed June 30, 2017.
- 5. ICH Harnomised Tripartite Guidelines. Statistical Principles for Clinical Trials. 1998; http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E9/Step4/E9\_Guideline.pdf. Accessed June 30, 2017.
- 6. Chan AW, Tetzlaff JM, Altman DG, et al. SPIRIT 2013 statement: defining standard protocol items for clinical trials. *Ann Intern Med.* 2013;158(3):200-207.
- 7. Chan AW, Tetzlaff JM, Gotzsche PC, et al. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. *BMJ*. 2013;346:e7586.
- 8. Merchant RM, Yang L, Becker LB, et al. Incidence of treated cardiac arrest in hospitalized patients in the United States. *Crit Care Med.* 2011;39(11):2401-2406.
- 9. DANARREST sterring commitee. DANARREST Registrering af hjertestop på hospital. Årsrapport 2015 [Danish]. 2016; https://www.sundhed.dk/content/cms/83/70283\_danarrest-%C3%A5rsrapport-2015.pdf. Accessed 6/5, 2017.
- 10. Benjamin EJ, Blaha MJ, Chiuve SE, et al. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. *Circulation*. 2017;135(10):e146-e603.
- 11. Andersen LW, Granfeldt A, Callaway CW, et al. Association Between Tracheal Intubation During Adult In-Hospital Cardiac Arrest and Survival. *JAMA*. 2017;317(5):494-506.
- 12. Engsig M, Soholm H, Folke F, et al. Similar long-term survival of consecutive in-hospital and out-of-hospital cardiac arrest patients treated with targeted temperature management. *Clin Epidemiol*. 2016;8:761-768.

- 13. Chan PS, Nallamothu BK, Krumholz HM, et al. Long-term outcomes in elderly survivors of in-hospital cardiac arrest. *N Engl J Med.* 2013;368(11):1019-1026.
- 14. Chan PS, Nallamothu BK, Krumholz HM, et al. Readmission rates and long-term hospital costs among survivors of an in-hospital cardiac arrest. *Circ Cardiovasc Qual Outcomes*. 2014;7(6):889-895.
- 15. Ornato JP, Becker LB, Weisfeldt ML, Wright BA. Cardiac arrest and resuscitation: an opportunity to align research prioritization and public health need. *Circulation*. 2010;122(18):1876-1879.
- Coute R, Panchal A, Mader T, Neumar R. National Institutes of Health–Funded Cardiac Arrest
   Research: A 10-Year Trend Analysis. *Journal of the American Heart Association*. 2017;6(7):6:e005239.
- 17. Morrison LJ, Neumar RW, Zimmerman JL, et al. Strategies for improving survival after in-hospital cardiac arrest in the United States: 2013 consensus recommendations: a consensus statement from the American Heart Association. *Circulation*. 2013;127(14):1538-1563.
- 18. Sinha SS, Sukul D, Lazarus JJ, et al. Identifying Important Gaps in Randomized Controlled Trials of Adult Cardiac Arrest Treatments: A Systematic Review of the Published Literature. *Circ Cardiovasc Qual Outcomes*. 2016;9(6):749-756.
- 19. Hazinski MF, Nolan JP, Aickin R, et al. Part 1: Executive Summary: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. *Circulation*. 2015;132(16 Suppl 1):S2-39.
- Soar J, Nolan JP, Bottiger BW, et al. European Resuscitation Council Guidelines for Resuscitation
   2015: Section 3. Adult advanced life support. *Resuscitation*. 2015;95:100-147.
- 21. Link MS, Berkow LC, Kudenchuk PJ, et al. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015;132(18 Suppl 2):S444-464.
- Jacobs IG, Finn JC, Jelinek GA, Oxer HF, Thompson PL. Effect of adrenaline on survival in out-of-hospital cardiac arrest: A randomised double-blind placebo-controlled trial. *Resuscitation*.
   2011;82(9):1138-1143.
- 23. Kudenchuk PJ, Brown SP, Daya M, et al. Amiodarone, Lidocaine, or Placebo in Out-of-Hospital Cardiac Arrest. *N Engl J Med.* 2016;374(18):1711-1722.
- 24. Chan PS, Spertus JA, Krumholz HM, et al. A validated prediction tool for initial survivors of in-hospital cardiac arrest. *Arch Intern Med.* 2012;172(12):947-953.
- 25. Wang CH, Huang CH, Chang WT, et al. Monitoring of serum lactate level during cardiopulmonary resuscitation in adult in-hospital cardiac arrest. *Crit Care*. 2015;19:344.
- 26. Nolan JP, Neumar RW, Adrie C, et al. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A Scientific Statement from the International Liaison Committee on

- Resuscitation; the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; the Council on Stroke. *Resuscitation*. 2008;79(3):350-379.
- 27. Busl KM, Greer DM. Hypoxic-ischemic brain injury: pathophysiology, neuropathology and mechanisms. *NeuroRehabilitation*. 2010;26(1):5-13.
- 28. Chalkias A, Xanthos T. Post-cardiac arrest brain injury: pathophysiology and treatment. *J Neurol Sci.* 2012;315(1-2):1-8.
- 29. Trzeciak S, Jones AE, Kilgannon JH, et al. Significance of arterial hypotension after resuscitation from cardiac arrest. *Crit Care Med.* 2009;37(11):2895-2903; quiz 2904.
- 30. Mutlu GM, Factor P. Role of vasopressin in the management of septic shock. *Intensive Care Med.* 2004;30(7):1276-1291.
- 31. Delmas A, Leone M, Rousseau S, Albanese J, Martin C. Clinical review: Vasopressin and terlipressin in septic shock patients. *Crit Care*. 2005;9(2):212-222.
- 32. Baumann G, Dingman JF. Distribution, blood transport, and degradation of antidiuretic hormone in man. *J Clin Invest.* 1976;57(5):1109-1116.
- 33. Rhodes A, Evans LE, Alhazzani W, et al. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. *Crit Care Med.* 2017;45(3):486-552.
- 34. Cossu AP, Mura P, De Giudici LM, et al. Vasopressin in hemorrhagic shock: a systematic review and meta-analysis of randomized animal trials. *Biomed Res Int.* 2014;2014:421291.
- 35. Saner FH, Canbay A, Gerken G, Broelsch CE. Pharmacology, clinical efficacy and safety of terlipressin in esophageal varices bleeding, septic shock and hepatorenal syndrome. *Expert Rev Gastroenterol Hepatol.* 2007;1(2):207-217.
- 36. Rembratt A, Graugaard-Jensen C, Senderovitz T, Norgaard JP, Djurhuus JC. Pharmacokinetics and pharmacodynamics of desmopressin administered orally versus intravenously at daytime versus night-time in healthy men aged 55-70 years. *Eur J Clin Pharmacol*. 2004;60(6):397-402.
- 37. Lindner KH, Haak T, Keller A, Bothner U, Lurie KG. Release of endogenous vasopressors during and after cardiopulmonary resuscitation. *Heart.* 1996;75(2):145-150.
- 38. Miano TA, Crouch MA. Evolving role of vasopressin in the treatment of cardiac arrest. *Pharmacotherapy.* 2006;26(6):828-839.
- 39. Paradis NA, Martin GB, Rivers EP, et al. Coronary perfusion pressure and the return of spontaneous circulation in human cardiopulmonary resuscitation. *JAMA*. 1990;263(8):1106-1113.

- 40. Wenzel V, Krismer AC, Arntz HR, Sitter H, Stadlbauer KH, Lindner KH. A comparison of vasopressin and epinephrine for out-of-hospital cardiopulmonary resuscitation. *N Engl J Med.* 2004;350(2):105-113.
- 41. Mentzelopoulos SD, Zakynthinos SG, Siempos I, Malachias S, Ulmer H, Wenzel V. Vasopressin for cardiac arrest: meta-analysis of randomized controlled trials. *Resuscitation*. 2012;83(1):32-39.
- 42. Gueugniaud PY, David JS, Chanzy E, et al. Vasopressin and epinephrine vs. epinephrine alone in cardiopulmonary resuscitation. *N Engl J Med.* 2008;359(1):21-30.
- 43. Layek A, Maitra S, Pal S, Bhattacharjee S, Baidya DK. Efficacy of vasopressin during cardio-pulmonary resuscitation in adult patients: a meta-analysis. *Resuscitation*. 2014;85(7):855-863.
- 44. Stiell IG, Hebert PC, Wells GA, et al. Vasopressin versus epinephrine for inhospital cardiac arrest: a randomised controlled trial. *Lancet*. 2001;358(9276):105-109.
- 45. Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, et al. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. *Arch Intern Med.* 2009;169(1):15-24.
- 46. Mentzelopoulos SD, Malachias S, Chamos C, et al. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. *JAMA*. 2013;310(3):270-279.
- 47. Guyton AC, Hall JE. *Textbook of Medical Physiology*. 11th ed: Elsevier Inc.; 2006.
- 48. Sapolsky RM, Romero LM, Munck AU. How do glucocorticoids influence stress responses?

  Integrating permissive, suppressive, stimulatory, and preparative actions. *Endocr Rev.* 2000;21(1):55-89.
- 49. Stahn C, Lowenberg M, Hommes DW, Buttgereit F. Molecular mechanisms of glucocorticoid action and selective glucocorticoid receptor agonists. *Molecular and cellular endocrinology.* 2007;275(1-2):71-78.
- 50. Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. *Clin Pharmacokinet*. 2005;44(1):61-98.
- 51. Hafezi-Moghadam A, Simoncini T, Yang Z, et al. Acute cardiovascular protective effects of corticosteroids are mediated by non-transcriptional activation of endothelial nitric oxide synthase.

  Nat Med. 2002;8(5):473-479.
- 52. Hall ED. The neuroprotective pharmacology of methylprednisolone. *J Neurosurg.* 1992;76(1):13-22.
- 53. Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. *N Engl J Med.* 2005;353(16):1711-1723.

- 54. World Health Organization. WHO Model List of Essential Medicines 2015;
  http://www.who.int/medicines/publications/essentialmedicines/EML\_2015\_FINAL\_amended\_NOV2
  015.pdf?ua=1. Accessed July 18, 2017.
- 55. Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating sepsis.

  \*Cochrane Database Syst Rev. 2015(12):CD002243.
- 56. Lindner KH, Strohmenger HU, Ensinger H, Hetzel WD, Ahnefeld FW, Georgieff M. Stress hormone response during and after cardiopulmonary resuscitation. *Anesthesiology*. 1992;77(4):662-668.
- 57. Smithline H, Rivers E, Appleton T, Nowak R. Corticosteroid supplementation during cardiac arrest in rats. *Resuscitation*. 1993;25(3):257-264.
- 58. Shi WL, Zhang T, Zhou JR, Huang YH, Jiang CL. Rapid permissive action of dexamethasone on the regulation of blood pressure in a rat model of septic shock. *Biomed Pharmacother*. 2016;84:1119-1125.
- 59. Varvarousi G, Stefaniotou A, Varvaroussis D, Xanthos T. Glucocorticoids as an emerging pharmacologic agent for cardiopulmonary resuscitation. *Cardiovasc Drugs Ther.* 2014;28(5):477-488.
- 60. Botnaru T, Altherwi T, Dankoff J. Improved neurologic outcomes after cardiac arrest with combined administration of vasopressin, steroids, and epinephrine compared to epinephrine alone. *CJEM*. 2015;17(2):202-205.
- 61. Ballew KA. ACP Journal Club. Combined vasopressin, steroids, and epinephrine improved survival in in-hospital cardiac arrest. *Ann Intern Med.* 2013;159(10):JC4.
- 62. Buddineni JP, Callaway C, Huang DT. Epinephrine, vasopressin and steroids for in-hospital cardiac arrest: the right cocktail therapy? *Crit Care*. 2014;18(3):308.
- 63. Hwang JY, Arredondo AF, Paul TK. Lung cancer screening, targeted temperature after cardiac arrest, and vasopressin and steroids in cardiac arrest. *Am J Respir Crit Care Med.* 2014;189(8):994-995.
- 64. Donnino MW, Andersen LW, Berg KM, et al. Corticosteroid therapy in refractory shock following cardiac arrest: a randomized, double-blind, placebo-controlled, trial. *Crit Care.* 2016;20:82.
- 65. Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. *J Clin Epidemiol.* 1999;52(1):19-26.
- 66. Krag M, Perner A, Wetterslev J, et al. Stress ulcer prophylaxis with a proton pump inhibitor versus placebo in critically ill patients (SUP-ICU trial): study protocol for a randomised controlled trial.

  Trials. 2016;17(1):205.
- 67. Fergusson D, Aaron SD, Guyatt G, Hebert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. *BMJ*. 2002;325(7365):652-654.

- 68. Mhyre JM, Tsen LC, Einav S, Kuklina EV, Leffert LR, Bateman BT. Cardiac arrest during hospitalization for delivery in the United States, 1998-2011. *Anesthesiology*. 2014;120(4):810-818.
- 69. Jeejeebhoy FM, Zelop CM, Lipman S, et al. Cardiac Arrest in Pregnancy: A Scientific Statement From the American Heart Association. *Circulation*. 2015;132(18):1747-1773.
- 70. Nichol G, Powell JL, Emerson S. On coenrollment in clinical resuscitation studies: review and experience from randomized trials. *Resuscitation*. 2010;81(7):792-795.
- 71. Andersen LW. DANRREST Registrering af hjertestop på hospital. Dokumentalistrapport [Danish].

  2017; http://www.rkkp.dk/siteassets/om-rkkp/de-kliniskekvalitetsdatabaser/danarrest/dokumentalistrapport-danarrest-juli-2017-inkl-bilag.pdf. Accessed July
  13, 2017.
- 72. Cummins RO, Chamberlain D, Hazinski MF, et al. Recommended guidelines for reviewing, reporting, and conducting research on in-hospital resuscitation: the in-hospital 'Utstein style'. A statement for healthcare professionals from the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, the Australian Resuscitation Council, and the Resuscitation Councils of Southern Africa. *Resuscitation*. 1997;34(2):151-183.
- 73. Perkins GD, Jacobs IG, Nadkarni VM, et al. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: A Statement for Healthcare Professionals From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. *Resuscitation*. 2015;96:328-340.
- 74. Becker LB, Aufderheide TP, Geocadin RG, et al. Primary outcomes for resuscitation science studies: a consensus statement from the American Heart Association. *Circulation*. 2011;124(19):2158-2177.
- 75. Jennett B, Bond M. Assessment of outcome after severe brain damage. *Lancet.* 1975;1(7905):480-484.
- 76. Pouw ME, Peelen LM, Moons KG, Kalkman CJ, Lingsma HF. Including post-discharge mortality in calculation of hospital standardised mortality ratios: retrospective analysis of hospital episode statistics. *BMJ*. 2013;347:f5913.

- 77. Vasilevskis EE, Kuzniewicz MW, Dean ML, et al. Relationship between discharge practices and intensive care unit in-hospital mortality performance: evidence of a discharge bias. *Med Care*. 2009;47(7):803-812.
- 78. Drye EE, Normand SL, Wang Y, et al. Comparison of hospital risk-standardized mortality rates calculated by using in-hospital and 30-day models: an observational study with implications for hospital profiling. *Ann Intern Med.* 2012;156(1 Pt 1):19-26.
- 79. Schoenfeld DA, Bernard GR, ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. *Crit Care Med.* 2002;30(8):1772-1777.
- 80. Vincent JL, Moreno R, Takala J, et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. *Intensive Care Med.* 1996;22(7):707-710.
- 81. Brown SM, Duggal A, Hou PC, et al. Nonlinear Imputation of PaO2/FIO2 From SpO2/FIO2 Among Mechanically Ventilated Patients in the ICU: A Prospective, Observational Study. *Crit Care Med.* 2017.
- 82. Brown SM, Grissom CK, Moss M, et al. Nonlinear Imputation of Pao2/Fio2 From Spo2/Fio2 Among Patients With Acute Respiratory Distress Syndrome. *Chest.* 2016;150(2):307-313.
- 83. van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. *Stroke*. 1988;19(5):604-607.
- 84. Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. *J Neurotrauma*. 1998;15(8):573-585.
- 85. Schmidt M, Schmidt SA, Sandegaard JL, Ehrenstein V, Pedersen L, Sorensen HT. The Danish National Patient Registry: a review of content, data quality, and research potential. *Clin Epidemiol*. 2015;7:449-490.
- 86. Herdman M, Gudex C, Lloyd A, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). *Qual Life Res.* 2011;20(10):1727-1736.
- 87. McPhail S, Lane P, Russell T, et al. Telephone reliability of the Frenchay Activity Index and EQ-5D amongst older adults. *Health Qual Life Outcomes*. 2009;7:48.
- 88. Patel N, Rao VA, Heilman-Espinoza ER, Lai R, Quesada RA, Flint AC. Simple and reliable determination of the modified rankin scale score in neurosurgical and neurological patients: the mRS-9Q.

  Neurosurgery. 2012;71(5):971-975; discussion 975.

- 89. Haywood K, Whitehead L, Nadkarni VM, et al. COSCA (Core Outcome Set for Cardiac Arrest) in Adults: An Advisory Statement From the International Liaison Committee on Resuscitation. *Circulation*. 2018;137(22):e783-e801.
- 90. Larkin GL, Copes WS, Nathanson BH, Kaye W. Pre-resuscitation factors associated with mortality in 49,130 cases of in-hospital cardiac arrest: a report from the National Registry for Cardiopulmonary Resuscitation. *Resuscitation*. 2010;81(3):302-311.
- 91. Morgan RW, Fitzgerald JC, Weiss SL, Nadkarni VM, Sutton RM, Berg RA. Sepsis-associated in-hospital cardiac arrest: Epidemiology, pathophysiology, and potential therapies. *J Crit Care*. 2017;40:128-135.
- 92. Tran S, Deacon N, Minokadeh A, et al. Frequency and survival pattern of in-hospital cardiac arrests:

  The impacts of etiology and timing. *Resuscitation*. 2016;107:13-18.
- 93. Bergum D, Nordseth T, Mjolstad OC, Skogvoll E, Haugen BO. Causes of in-hospital cardiac arrest incidences and rate of recognition. *Resuscitation*. 2015;87:63-68.
- 94. Wallmuller C, Meron G, Kurkciyan I, Schober A, Stratil P, Sterz F. Causes of in-hospital cardiac arrest and influence on outcome. *Resuscitation*. 2012;83(10):1206-1211.
- 95. Nolan JP, Soar J, Cariou A, et al. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. *Resuscitation*. 2015;95:202-222.
- 96. Lindner G, Funk GC. Hypernatremia in critically ill patients. J Crit Care. 2013;28(2):216 e211-220.
- 97. Brandt LJ, Feuerstadt P, Longstreth GF, Boley SJ, American College of G. ACG clinical guideline: epidemiology, risk factors, patterns of presentation, diagnosis, and management of colon ischemia (CI). *Am J Gastroenterol.* 2015;110(1):18-44; quiz 45.
- 98. Singer M, Deutschman CS, Seymour CW, et al. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). *JAMA*. 2016;315(8):801-810.
- 99. Shankar-Hari M, Phillips GS, Levy ML, et al. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). *JAMA*. 2016;315(8):775-787.
- 100. Seymour CW, Liu VX, Iwashyna TJ, et al. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). *JAMA*. 2016;315(8):762-774.
- 101. Tsai MS, Chiang WC, Lee CC, et al. Infections in the survivors of out-of-hospital cardiac arrest in the first 7 days. *Intensive Care Med.* 2005;31(5):621-626.
- 102. Mongardon N, Perbet S, Lemiale V, et al. Infectious complications in out-of-hospital cardiac arrest patients in the therapeutic hypothermia era. *Crit Care Med.* 2011;39(6):1359-1364.

- 103. Gagnon DJ, Nielsen N, Fraser GL, et al. Prophylactic antibiotics are associated with a lower incidence of pneumonia in cardiac arrest survivors treated with targeted temperature management.

  \*Resuscitation. 2015;92:154-159.
- 104. Kalanuria AA, Ziai W, Mirski M. Ventilator-associated pneumonia in the ICU. *Crit Care*. 2014;18(2):208.
- 105. Laupland KB, Bagshaw SM, Gregson DB, Kirkpatrick AW, Ross T, Church DL. Intensive care unit-acquired urinary tract infections in a regional critical care system. *Crit Care*. 2005;9(2):R60-65.
- 106. Goldberger ZD, Chan PS, Berg RA, et al. Duration of resuscitation efforts and survival after in-hospital cardiac arrest: an observational study. *Lancet*. 2012;380(9852):1473-1481.
- 107. Schulz KF, Altman DG, Moher D, Group C. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. *BMJ*. 2010;340:c332.
- 108. Moher D, Hopewell S, Schulz KF, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. *BMJ*. 2010;340:c869.
- 109. Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med. 1985;4(2):213-226.
- 110. Fernando SM, Tran A, Cheng W, et al. Pre-arrest and intra-arrest prognostic factors associated with survival after in-hospital cardiac arrest: systematic review and meta-analysis. *BMJ*. 2019;367:l6373.
- 111. Hernandez AV, Steyerberg EW, Habbema JD. Covariate adjustment in randomized controlled trials with dichotomous outcomes increases statistical power and reduces sample size requirements. *J Clin Epidemiol.* 2004;57(5):454-460.
- 112. Kahan BC, Jairath V, Dore CJ, Morris TP. The risks and rewards of covariate adjustment in randomized trials: an assessment of 12 outcomes from 8 studies. *Trials*. 2014;15:139.
- 113. Kahan BC. Accounting for centre-effects in multicentre trials with a binary outcome when, why, and how? *BMC Med Res Methodol*. 2014;14:20.
- 114. Spiegelman D, Hertzmark E. Easy SAS calculations for risk or prevalence ratios and differences. *Am J Epidemiol.* 2005;162(3):199-200.
- 20u G. A modified poisson regression approach to prospective studies with binary data. *Am J Epidemiol.* 2004;159(7):702-706.
- 116. Mantel N. Chi-square test with one degreee of freedom: Extension of the Mantel-Haenszel Procedure *Journal of the American Statistical Association*. 1963;58(303):690-700.
- 117. Kahan BC, Morris TP. Reporting and analysis of trials using stratified randomisation in leading medical journals: review and reanalysis. *BMJ*. 2012;345:e5840.
- 118. Kaufman JS, MacLehose RF. Which of these things is not like the others? *Cancer.* 2013;119(24):4216-4222.

- 119. Assmann SF, Pocock SJ, Enos LE, Kasten LE. Subgroup analysis and other (mis)uses of baseline data in clinical trials. *Lancet*. 2000;355(9209):1064-1069.
- 120. van Elteren P. On the Combination of Independent Two Sample Tests of Wilcoxon. *Bulletin of the Institute of International Statistics*. 1960;37:351-361.
- 121. Fleming T, Harrington D. Nonparametric estimation of the survival distribution in censored data.

  \*Communications in Statistics Theory and Methods. 1984;13(20):2469–2486.
- 122. Cox D. Regression models and life tables. *Journal of the Royal Statistical Society*. 1972; Series B(20):187–220.
- 123. Kleinbaum D, Klein M. Survival Analysis: A Self-Learning Text. 3rd ed: Springer; 2013.
- 124. McCullagh P. Regression Models for Ordinal Data. *Journal of the Royal Statistical Society*. 1980;42(2):109-142.
- 125. Rothman KJ. No Adjustments Are Needed for Multiple Comparisons. *Epidemiology.* 1990;1(1):43-46.
- 126. Feise RJ. Do multiple outcome measures require p-value adjustment? *BMC Med Res Methodol.* 2002;2:8.
- 127. Gibson D, Harvey AJ, Everett V, Parmar MK. Is double data entry necessary? The CHART trials. CHART Steering Committee. Continuous, Hyperfractionated, Accelerated Radiotherapy. *Control Clin Trials*. 1994;15(6):482-488.
- 128. Day S, Fayers P, Harvey D. Double data entry: what value, what price? *Control Clin Trials*. 1998;19(1):15-24.
- 129. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. *J Biomed Inform*. 2009;42(2):377-381.
- 130. Monsieurs KG, Nolan JP, Bossaert LL, et al. European Resuscitation Council Guidelines for Resuscitation 2015: Section 1. Executive summary. *Resuscitation*. 2015;95:1-80.
- 131. Danish Resuscitation Council. Advanced resusciation [Danish]. http://genoplivning.dk/avanceret-genoplivning/.
- 132. Bossaert LL, Perkins GD, Askitopoulou H, et al. European Resuscitation Council Guidelines for Resuscitation 2015: Section 11. The ethics of resuscitation and end-of-life decisions. *Resuscitation*. 2015;95:302-311.
- 133. Annane D. What Is the Evidence for Harm of Neuromuscular Blockade and Corticosteroid Use in the Intensive Care Unit? *Semin Respir Crit Care Med.* 2016;37(1):51-56.
- 134. Annane D, Bellissant E, Bollaert PE, et al. Corticosteroids in the treatment of severe sepsis and septic shock in adults: a systematic review. *JAMA*. 2009;301(22):2362-2375.

- 135. Bulkley BH, Roberts WC. Steroid therapy during acute myocardial infarction. A cause of delayed healing and of ventricular aneurysm. *Am J Med.* 1974;56(2):244-250.
- 136. Giugliano GR, Giugliano RP, Gibson CM, Kuntz RE. Meta-analysis of corticosteroid treatment in acute myocardial infarction. *Am J Cardiol*. 2003;91(9):1055-1059.
- 137. van Belle G, Mentzelopoulos SD, Aufderheide T, May S, Nichol G. International variation in policies and practices related to informed consent in acute cardiovascular research: Results from a 44 country survey. *Resuscitation*. 2015;91:76-83.
- 138. Mentzelopoulos SD, Mantzanas M, van Belle G, Nichol G. Evolution of European Union legislation on emergency research. *Resuscitation*. 2015;91:84-91.
- 139. Lov om videnskabsetisk behandling af sundhedsvidenskabelige forskningsprojekter [Danish]. 2011; https://www.retsinformation.dk/forms/r0710.aspx?id=137674#Not1. Accessed July 7, 2017.
- 140. Vejledning om akutte forsøg [Danish]. 2017; http://www.nvk.dk/emner/akutte-forsoeg/vejledning-om-akutte-forsoeg#1. Accessed July 7, 2017.
- 141. Lov om kliniske forsøg med lægemidler [Danish]. 2016; https://www.retsinformation.dk/Forms/r0710.aspx?id=180117. Accessed July 7, 2017.
- 142. Vognsen M, Fabian-Jessing BK, Secher N, et al. Contemporary animal models of cardiac arrest: A systematic review. *Resuscitation*. 2017;113:115-123.
- 143. Donnino MW, Salciccioli JD, Howell MD, et al. Time to administration of epinephrine and outcome after in-hospital cardiac arrest with non-shockable rhythms: retrospective analysis of large in-hospital data registry. *BMJ*. 2014;348:g3028.
- 144. Ministeriet for Sundhed og Forebyggelse. Letter to Den Nationale Videnskabsetiske Komité dated February 28th, 2014 regarding "Anvendelse af data i akutforsøg" [Danish]. In.
- 145. Lov om ændring af lov om videnskabsetisk behandling af sundhedsvidenskabelige forskningsprojekter [Danish]. 2012; https://www.retsinformation.dk/forms/r0710.aspx?id=142351. Accessed July 13, 2017.
- 146. Bekendtgørelse af lov om klage- og erstatningsadgang inden for sundhedsvæsenet [Danish]. 2011; https://www.retsinformation.dk/Forms/r0710.aspx?id=138893. Accessed July 13, 2017.
- 147. International Committee of Medical Journal Editors. Defining the Role of Authors and Contributors.
  2017; http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html. Accessed July 6, 2017.
- 148. Taichman DB, Sahni P, Pinborg A, et al. Data Sharing Statements for Clinical Trials A Requirement of the International Committee of Medical Journal Editors. *N Engl J Med.* 2017;376(23):2277-2279.

# **Appendices**

## Appendix 1: Conflict of interest disclosures for the steering committee members

#### Lars W. Andersen

None

#### Other:

- Member of the Advanced Life Support task force at ILCOR
- Editorial board member at Resuscitation
- Member of the steering committee at DANARREST
- Honorarium from JAMA for statistical reviews

## **Hans Kirkegaard**

#### Industry:

• None

#### Other:

• Chairman of the steering committee for DANARREST

## **Michael Donnino**

#### Industry:

• Research grants from Kaneka, General Electric, and Bristol-Myers-Squibb

## Other:

- Research grants from the American Heart Association and the National Institute of Health
- Vice-chair of the Advanced Life Support task force at ILCOR

## **Tobias Kurth**

## Industry:

Lecture fees from Novartis

Other:

Honorarium from the BMJ for editorial services **Bodil S. Rasmussen** Industry: Research grant from Ferring Other: None Jesper Kjærgaard Industry: Lecture fees from Orion Pharma, AstraZeneca, and Bayer Other: None Bo Løfgren Industry: Lecture fees from Boehringer Ingelheim, AstraZeneca, and Bayer Recipient of a teaching award from the Danish Society of Cardiology sponsored by Merck Sharp and Dohme Other: Member of The European Resuscitation Council Basic Life Support and Automated External Defibrillation International Course Committee (2010 – 2016) Member of the Basic Life Support task force at ILCOR (2017 – 2020) **Asger Granfeldt** Industry: None Other:

None

| Industry: |
|-------------------------|
| • None |
| Other: |
| • None |
| Stine Thorhauge Zwisler |
| Industry: |
| • None |
| Other: |
| None |
| Søren Darling |
| Industry: |
| None |
| Other: |
| None |
| Kasper Glerup Lauridsen |
| Industry: |
| None |

Jacob Moesgaard Larsen Industry:

None

None

Other:

Dan Isbye

| <ul> <li>European Resuscitation Council Advanced Life Support (ALS) Science and Educational Committee member.</li> <li>Kim B. Pælestik</li> <li>Industry: <ul> <li>None</li> </ul> </li> <li>Other: <ul> <li>None</li> </ul> </li> <li>Christoffer Sølling</li> </ul> <li>Industry: <ul> <li>Industry:</li> <li>Industry:</li> <li>Industry:</li> </ul> </li> | r: |
|---|---|
| Kim B. Pælestik Industry: • None Other: • None Christoffer Sølling Industry: | European Resuscitation Council Advanced Life Support (ALS) Science and Educational Committee |
| Industry: None Other: None Christoffer Sølling Industry: | member. |
| Industry: None Other: None Christoffer Sølling Industry: | |
| <ul> <li>None</li> <li>Other: <ul> <li>None</li> </ul> </li> <li>Christoffer Sølling</li> <li>Industry:</li> </ul> | B. Pælestik |
| Other: • None Christoffer Sølling Industry: | stry: |
| None Christoffer Sølling Industry: | None |
| None Christoffer Sølling Industry: | |
| Christoffer Sølling Industry: | r: |
| Industry: | None |
| Industry: | |
| | toffer Sølling |
| •• | stry: |
| • None | None None |
| Other: | r: |
| • None | None |
| Anders Kjærgaard | |
| Industry: | |
| • None | None |
| Other: | |
| • None | None |
| Dorte Due-Rasmussen | o Duo Parmurran |
| Industry: | |
| • None | None |
| Other: | ٠٠, |
| None | |

| Industry | <b>':</b> |
|-----------|-------------|
| • 1 | None |
| Other: | |
| • | None |
| Fredrik I | Folke |
| Industry | : |
| • 1 | None |
| Other: | |
| | None |
| Mette G | itz Charlot |
| Industry | <b>:</b> : |
| • | None |
| Other: | |
| • | None |
| Sebastia | an Wiberg |
| Industry | ·: |
| • | None |

**Kasper Iversen** 

None

• None

**Martin Schultz** 

Industry:

Other:

| Other: | |
|---------|-------------|
| • | None |
| Mathia | as Holmberg |
| Industr | ry: |
| • | None |
| Other: | |
| • | None |

Other:

Industry:

• None

• None

Rikke Malene Jepsen

# Appendix 2: Study kit and drug labeling (Danish)

Example from the Aarhus site.



| vares ved mellem 2 og 8 °C.<br>og maksimalt til angivet |
|---|
| g maksimalt til angivet |
| g maksimalt til angivet |
| - |
| Afblinding: Ved alvorlig bivirkning som kan formodes at skyldes |
| studiemedicin kan afblinding foretages vha. kuverten i bunden af æsken. |
| Kuverten skal lægges tilbage i æsken efter brug. |
| Æsken: ROSC: Æsken skal følge patienten. |
| sansvarlige. |
| r |

Fremstillet af Skanderborg Apotek

## Α

#### Solu-Medrol/placebo **SOLVENS 1ml**

til opl. til injektion 1ml Randomiseringsnr. XXXX Anv. Inden 00-0000 Batchnr. 0000 VAM-IHCA

## В

#### Solu-Medrol/placebo **PULVER**

til opl.til i.v. injektion 40mg Randomiseringsnr. XXXX Anv. Inden 00-0000 Batchnr. 0000 VAM-IHCA

# C

#### Empressin/placebo

til i.v. adm. 2ml Randomiseringsnr. XXXX Randomiseringsnr. XXXX Anv. Inden 00-0000 Batchnr. 0000 VAM-IHCA

## Appendix 3: Draft of CONSORT flow diagram



# Appendix 4: Case report form (Danish)

# REGISTRERINGSSKEMA - VAM-IHCA

Randomiseringsnummer: \_\_\_\_\_

| 1) Patientnavn og CPR-nr.: | 2) Skema udfyldt af: |
|---|---|
| Navn: | Navn: |
| CPR: | Arbejdsmail: |
| 3) Dato og tid for konstatering af | 4) Studiemedicin givet: |
| hjertestoppet: | |
| DD MM Å Å | JA NEJ → Årsag: |
| Dato: / / | |
| | ROSC |
| T T M M | Udfyld resten Ingen IV/IO |
| Tid: : | af skemaet Andet: |
| 5) Tid for første adrenalin administration: | 6) Tid for første vasopressin/placebo |
| | (ampul C + C) administration: |
| T T M M | T T M M |
| Tid: | Tid: |
| 7) Methylprednisolon/placebo | 8) Total antal vasopressin/placebo |
| (hætteglas A + B) administreret? | (ampul C + C) administreret: |
| maccegias A + b) duministrerect | |
| JA NEJ | 1 2 3 4 |
| JA NE | |
| 9) ROSC (egencirkulation) opnået? | ROSC: Return Of Spontaneus Circulation |
| 5, 11000 (egenerikalation) opnacti | (egencirkulation) defineres som spontan |
| JA NEJ ECMO/CPB | cirkulation (dvs. en mærkbar puls eller måleligt |
| za les comojers | blodtryk) uden yderligere behov for hjertemassage, |
| | der opretholdes i mindst 20 minutter. |

Ved ROSC følger medicinæsken, med indhold og registreringsskema, patienten. Hvis ROSC ikke opnås, medbringes æsken af den forsøgsansvarlige.

Husk endvidere venligst at udfylde DANARREST.

Evt. noter eller kommentarer kan tilføjes på bagsiden.

Ved spørgsmål:

Mobil nr.: 93 52 10 42 (døgnet rundt)

E-mail: hjertestop@clin.au.dk

Registreringsskema v. 1.2 VAM-IHCA

# Appendix 5: DANARREST case report form (Danish)

| VEJLEDNING:<br>SE BAGSIDEN DANARREST – registr | rering af hjertestop på hospital |
|---|---|
| Patientnavn + CPR-nr. (evt. label) Navn: CPR-nr: | 2 Skema udfyldt af: Navn: Tlf./kode: DATO: D |
| 3 Lokalitet Skadestue/modtagelse: Ambulatorium: Sengeafdeling: Operationsgang: Opvågningsafdeling: Intensiv afdeling: Kardiologisk laboratorium Andet: | Stophold alarmeret Hvis "Ja": KL: T T: M M DATO: D D M M A Å 1. Klinisk hjertestop 2. Klinisk hjertestop: Indikation for genoplivning Ja Nej Hvis "Nej " i "1" eller "2" udfyldes resten af skemaet IKKE |
| Blev hjertestoppets indtræden observeret Ja ☐ af sundhedspersonale ☐ af lægmand Nej ☐ Hjerterytmeovervåget hjertestop Ja ☐ Nej ☐ | 14 Tid for konstatering af hjertestop KL: TTT: MMM |
| Hjertestop erkendt af Sundhedspersonale Lægmand | Ingen KL: I I I I I I I I I I I I I I I I I I I |
| Basal genoplivning for Stopholdets ankomst Hjertemassage Ingen Ventilation Hjertemassage og ventilation Stophold ikke alarmeret | 17 Tid for <i>første</i> defibrillering KL: |
| Rytmeanalyse og defibrillering <b>før</b> Stopholdets ankomst Første hjerterytme Ikke-stødbar rytme Stødbar rytme Manuel defibrillator Defibrillering med Stophold ikke alarmeret | 18 Tid for Stopholdets ankomst KL: T T: M M Stophold ikke alarmeret 19 Genoplivning indstillet pga. Spontant kredsløb Død Død Kunstigt kredsløb (f.eks. ECMO, CPS, m.fl) KL: T T: M M DATO: D D / M M / Å Å |
| Den første observerede hjerterytme VF Pulsløs VT PEA Asystoli Ingen manuel rytmeanalyse Pulsgivende | 20 Årsag til hjertestop Non-kardial Formodet kardial |
| 1 1 Patientens status ved Stopholdets ankomst Hjertestop Ja Nej Nej Stophold ikke alarmeret 1 2 Medicin givet Adrenalin Amiodaron Ingen Andet: | Teammedlemmer/personale på Stopholdet |
| 13 Mekanisk hjertemassage Ja Nej | 22 Eventuelle kommentarer |

Version 3.0 (Rev. september 2016)

#### Vejledning til udfyldelse af registreringsskema

Registrering af hjertestop er vigtig for at dokumentere og forbedre behandlingen. Stopholdet er derfor som helhed ansvarlig for udfyldelse af skemaet. Skemaet udfyldes af lederen af Stopholdet, evt. med assistance fra et medlem af Stopholdet. Hvis Stopholdet ikke bliver tilkaldt, f.eks. på intensiv afdeling, operationsgang eller kardiologisk laboratorium, udfyldes skemaet af den for genoplivningen ansvarlige læge.

#### ALLE TIDSPUNKTER ANGIVES EFTER BEDSTE SKØN

- 1. Anfør patientnavn og CPR-nr. eller påsæt label.
- Anfør navn og telefon/personsøger på den person der har udfyldt skemaet. Angiv endvidere tidspunkt (dag, måned, år) for udfyldelse af skemaet.
- 3. Afkryds lokalitet, hvor hjertestoppet er indtrådt. Herudover anføres navn på lokaliteten. Ved kryds i "Andet" anføres lokalitet.
- Angiv tidspunkt (time, minut, dag, måned, år,) for hvornår Stopholdet alarmeres. Det tidspunkt der anføres, er det, hvor Omstillingen eller andet personale videreformidler alarmeringen til Stopholdet. Hvis Stophold ikke tilkaldes, sættes kryds i "Nej" og tidspunkt udfyldes ikke.
- 5. Skemaet skal udfyldes til <u>alle patienter med hjertestop på hospital, og til alle patienter hvor Stopholdet tilkaldes.</u> Skemaet skal således også udfyldes i fald patienten er blevet genopiivet INDEN Stopholdets ankomst. I fald patienten IKKE har eller har haft hjertestop ved Stopholdets ankomst eller der ikke er indikation for genopiivning, udfyldes kun punkt 1-5. Hvis en patient er genopiivet efter hjertestop uden for hospital (= ROSC> 20 min.), men får nyt hjertestop efter ankomst til hospital, skal skemaet ligeledes udfyldes. Der skal udfyldes et nyt skema, hvis en patient får et nyt hjertestop efter ROSC > 20 min. Hvis der forud for hjertestop foreligger en beslutning om "ingen genoplivning" afkrydses "Nej" i punkt 2. Hjertestop hos terminale patienter, hvor dødens indtræden forventes og hjertestopberedskabet ikke aktiveres, skal ikke registreres.
- Afkryds hvorvidt hjertestop er observeret af sundhedspersonale, lægmand eller er ubevidnet. "Observeret" indebærer, at man har set eller hørt personen få hjertestop, eller identificeret ventrikelflimmer på EKG-overvågning. Afkryds hvorvidt hjertestoppet var hjerterytmeovervåget. Med hjerterytmeovervåget menes monitoreret med EKG-overvågning (telemetri eller lignende).
- Afkryds hvorvidt hjertestoppet er erkendt af sundhedspersonale eller af lægmand. Erkendelsen af hjertestop beror på bevidstigshed og ikke normal vejrtrækning. For den trænede og erfarne behandler indgår pulsløshed ligeledes i diagnosen.
- Afkryds hvilken form for hjertelungeredning, der er ydet f\u00far Stopholdets ankomst. Hvis Stophold ikke tilkaldes, afkryds "Stophold ikke alarmeret", og undlad at udfylde den \u00favrige del af punktet.
- 9. Hjerterytmeanalyse før Stopholdets ankomst: Afkryds hvorvidt det drejer som en stødbar rytme, en ikke-stødbar rytme eller der ingen hjerterytmeanalyse er udført. Anvendes en AED, oplyses om der er stødbar rytme eller ikke-stødbar rytme. Ved brug af manuel defibrillator aflæses rytmen på apparatets skærm. Afkryds med hvilket apparatur rytmeanalyse er foretaget. Afkryds om der er foretaget defibrillering før Stopholdets ankomst (med AED eller manuelt) eller om der ingen defibrillering er foretaget. Hvis Stophold ikke tilkaldes, afkryds "Stophold ikke alarmeret", men øvrige punkter udfyldes.
- 10. Afkryds den først observerede hjerterytme relateret til hjertestop, uanset om denne er observeret af afdelingens personale eller af Stopholdet. Er der ikke gjort manuel rytmeanalyse ved at vurdere hjerterytmen på EKG-overvågning eller med manuel defibrillator afkrydses" Ingen manuel rytmeanalyse".
- Afkryds hvorvidt patienten har klinisk hjertestop ved Stopholdets ankomst. Hvis Stophold ikke tilkaldes, afkryds "Stophold ikke alarmeret", og undlad at udfylde den øvrige del af punktet.
- Afkryds hvilken medicin der er givet (sæt om nødvendigt flere krydser). Ved kryds i "Andet" anføres de anvendte farmaka på skemaet, f.eks. calciumchlorid, magnesiumsulfat, natriumbikarbonat, lidocain, mv.
- 13. Afkryds om der er givet mekanisk hjertemassage (f.eks. LUCAS® eller Autopulse®), om patienten var intuberet inden hjertestoppet eller om det er sket i forbindelse med hjertestopbehandlingen, og om der er anvendt kapnografi.
- 14. Angiv tidspunkt for konstatering af hjertestop (time, minut).
- 15. Angiv tidspunkt for påbegyndt hjertemassage eller ventilation (time, minut).
- 16. Angiv tidspunkt for første hjerterytmeanalyse (time, minut) (hjerterytmeanalyse med AED eller manuel defibrillator).
- 17. Angiv tidspunkt for første defibrillering (time, minut).
- Anfør tidspunkt for Stopholdets ankomst (time, minut). Hvis Stophold ikke tilkaldes, afkryds "Stophold ikke alarmeret", og undlad at udfylde den øvrige del af punktet. Ankomst af Stopholdet defineres ved ankomsten af lederen af Stopholdet.
- 19. Afkryds om genoplivningen er indstillet grundet genvundet spontant kredsløb, etablering af kunstigt kredsløb (ekstrakorporal cirkulation eller tilsvarende) eller om yderligere forsøg på genoplivning vurderes udsigtsløs ("Død"). Angiv tidspunkt (time, minut, dag, måned, år).
- Afkryds om der er en oplagt ikke-kardial årsag til hjertestoppet (f.eks. traumatisk, hypoxisk, forgiftning, drukning/hængning), og hvis det ikke er tilfældet – er årsagen formodet kardial.
- Personnavne eller personhenførbare data indtastes ikke i DANARREST, men anføres på papirskemaet (til opfølgning, debriefing o.lign). Den enkelte region/institution tager stilling til lokal praksis
- 22. Anfør eventuelle kommentarer til genoplivningsforløbet.

| Definitioner Stophold = hospitalets udrykningshold til behandling af hjertestop | Aflevering af udfyldte skemaer |
|---|---|
| Sundhedspersonale = læge, sygeplejerske, social- og sundhedsassistent, fysio-<br>og ergoterapeut, serviceassistent og portør | |
| Stødbar rytme – Ventrikelflimren og pulsløs ventrikulær takykardi<br>ikke-stødbar rytme – Asystoli og pulsløs elektrisk aktivitet | |
| VF = Ventrikelflimren Pulsiøs VT = Pulsiøs ventrikulær takykardi | |
| PEA = Pulsips elektrisk aktivitet<br>AED = Automatisk Ekstern Defibrillator ("Hjertestarter") | |

# Appendix 6: Charter for the independent data-monitoring committee (IDMC)

# Charter for the independent data-monitoring committee (IDMC) for the VAM-IHCA trial

**Trial name**: Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest – A Randomized, Double-Blind, Placebo-Controlled Trial (VAM-IHCA)

Principal investigator and sponsor: Associate professor Lars W. Andersen, M.D., M.P.H., Ph.D.

EudraCT Number: 2017-004773-13

Research ethical committee no.: 1-10-72-42-18, Central Denmark Region

#### Introduction

This charter will define the primary responsibilities of the IDMC, its relationship with other trial components, its membership, and the purpose and timing of its meetings. The charter will also provide the procedures for ensuring confidentiality and proper communication, the statistical monitoring guidelines to be implemented by the IDMC, and an outline of the content of the data that will be provided to the IDMC.

## Responsibilities of the IDMC

The IDMC will be responsible for safeguarding the interests of trial participants, assessing the safety and efficacy of the interventions during the trial, and for monitoring the overall conduct of the clinical trial. The IDMC will provide recommendations about stopping or continuing the trial to the steering committee of the VAM-IHCA trial. To contribute to enhancing the integrity of the trial, the IDMC may decide to also formulate recommendations relating to the selection/recruitment/retention of participants, their management, improving adherence to protocol-specified regimens and retention of participants, and the procedures for data management and quality control. Any such recommendations will be at the discretion of the IDMC.

The IDMC will be advisory to the steering committee. The steering committee will be responsible for promptly reviewing the IDMC recommendations, to decide whether to continue or terminate the trial, and to determine whether amendments to the protocol or changes in trial conduct are required.

The IDMC will be notified of all changes to the trial protocol or conduct. The IDMC concurrence will be sought on all substantive recommendations or changes to the protocol or trial conduct prior to their implementation.

The members of the IDMC will be unpaid.

#### Members of the IDMC

The IDMC is an independent multidisciplinary group consisting of physicians with epidemiological expertise that, collectively, has experience in the management of cardiac arrest patients and in the conduct, monitoring and analysis of randomized clinical trials.

The members of the IDMC are:

Christian Fynbo Christiansen, M.D., Ph.D. (chairman)

Clinical Associate Professor

Department of Clinical Epidemiology

Department of Clinical Medicine

Aarhus University, Aarhus, Denmark

Hans Friberg, M.D., Ph.D.

Professor

**Department of Clinical Sciences** 

Lund University, Lund, Sweden

&

Department of Perioperative and Intensive Care

Skåne University Hospital, Lund, Sweden

Jasmeet Soar, FRCA, FFICM, FRCP

Consultant

Anaesthesia and Intensive Care Medicine

Southmead Hospital, Bristol, United Kingdom

**Conflicts of interest** 

IDMC membership has been restricted to individuals free of conflicts of interest. The source of

these conflicts may be financial, scientific, or regulatory in nature. The IDMC members will disclose to fellow

members any consulting agreements or financial interests they have with the sponsor of the trial or with

other sponsors having products that are being evaluated or having products that are competitive with those

being evaluated in the trial. The IDMC will be responsible for deciding whether these consulting agreements

or financial interests materially impact their objectivity. The IDMC members will be responsible for advising

fellow members of any changes in these consulting agreements and financial interests that occur during the

trial. Any IDMC members who develop significant conflicts of interest during the trial should resign from the

IDMC.

IDMC membership is to be for the duration of the clinical trial. If any members leave the IDMC

during the trial, the steering committee will appoint the replacement(s).

VAM-IHCA Protocol - version 1.8

#### **Evaluations of trial data**

The IDMC will review deidentified data after six months of patient enrollment and then on a yearly basis (or more often if determined by the IDMC) for safety; unless there are group differences necessitating unblinding (as determined by the IDMC), the IDMC will be blinded to treatment groups. The trial will continue while the IDMC review data. After the review, the IDMC will create a short report to the steering committee with recommendations for continuation, modifications, or termination of the trial. There will be no formal stopping criteria for efficacy or futility. Criteria for recommending termination will be at the discretion of the IDMC and there will be no formal statistical criteria for termination due to safety.

Raw data will be provided to the IDMC in Excel in the following format:

Row 1 contains the names of the variables (to be defined below)

Row 2 to N (where N-1 is the number of patients who have entered the trial) each contains the data of one patient

Column 1 to p (where p is the number of variables to be defined below) each contains in row 1 the name of a variable and in the next N-1 rows the values of this variable.

The values of the following variables will be included:

1: id: a number that uniquely identifies the patient.

2: group: The randomization code (group A or B)

3: rosc: The primary outcome return of spontaneous circulation (ROSC) (1 for ROSC, 0 for no ROSC)

4: surv\_30: Survival at 30 days (1 for survival at 30 days, 0 for death prior to 30 days)

5: cpc\_30: Cerebral performance category (CPC) at hospital discharge (1 to 5)

Specific adverse events (see section 5.4.3 in the protocol):

6: hyp gly: Hyperglycemia (1 for yes, 0 for no)

7: insulin: Requirement for an insulin infusion (1 for yes, 0 for no)

8: Hyp na: Hypernatremia (1 for yes, 0 for no)

9: infect: New infections (1 for yes, 0 for no)

10: antibio: New or changing antibiotics (1 for yes, 0 for no)

11: gas bleed: Gastrointestinal bleeding (1 for yes, 0 for no)

12: mes ischemia: Mesenteric ischemia (1 for yes, 0 for no)

13: per\_ ischemia: Peripheral ischemia (1 for yes, 0 for no)

14: susar: Suspected Unexpected Serious Adverse Reactions (1 for yes, 0 for no)

Variables #1 and #3-14 will be provided by the steering committee and item #2 will be provided by the pharmacy.

An independent biostatistician (not a member of the IDMC) will provide aggregate data for each of the variables #3-12 stratified by treatment group (variable #2) in two-by-two tables. No statistical tests will be performed unless explicitly requested by the IDMC.

In addition to the above, the steering committee will provide the IDMC with data on the number of patients screened (i.e. all IHCA at participating sites), number of patients included in the studies, and the number of patients who have provided consent for additional data collection and long-term follow-up. Data will be provided on the specific reasons for non-inclusion and exclusion.

All data will be provided to the IDMC at least 5 days prior to their meeting.

#### Meeting, communication and reports

The steering committee, along with the IDMC chairman, will be responsible for scheduling and arranging the IDCM meeting. The meeting will start with a study overview provided by the principal investigator. This will include an overview of recruitment and potential problems and issues. The remainder of the meeting, which will only be attended by the IDMC members, be will be related to evaluations of trial data as described above.

The IDMC is not planned to meet physically to evaluate data. In addition to the scheduled meeting, the IDMC may whenever they decide, contact each other by telephone, videoconference, or e-mail to discuss the safety for trial participants. The recommendations of the IDMC regarding stopping, continuing or changing the design of the trial should be communicated in writing without delay to the steering committee. The steering committee has the responsibility to inform as fast as possible, and no later than 72 hours, all investigators of the trial and the sites including patients in the trial about the recommendation of the IDMC and the steering committee decision hereof.

The IDMC will prepare minutes of their meetings. The closed minutes will describe the

proceedings from all sessions of the IDMC meeting, including the listing of recommendations by the committee. Because it is possible that these minutes may contain unblinded information, it is important that they are not made available to anyone outside the IDMC. The IDMC and the independent biostatistician are obligated to keep all patient-level data confidential.